| iiaial Titla. Phaga II atudu of firat line treatment of Chronic Croft versus Heat Diag | |
|---|---|
| <b>icial Title:</b> Phase II study of first line treatment of Chronic Graft versus Host Dise | ase |
| h Arsenic Trioxide | |

**NCT Number:** 02966301

**Document Dates: SAP Amendment /** Version 3: 2020/12/21



Version 3.0 Date 21/12/2020

# STATISTICAL ANALYSIS PLAN

| Protocol Title: | Phase II study of first line treatment of Chronic Graft versus Host Disease with Arsenic Trioxide |
|---|---|
| Protocol | GMED16-001 |
| Number: | Eudract number: 2016-002358-18 |
| Compound: | ATO® |
| Phase: | Phase II |
| Sponsor: | MEDSENIC |
| | 204, avenue de Colmar |
| | F-67100 - Strasbourg |
| SAP Author: | Marine RAGOT-BENSEGHIR |
| SAP Version: | Version 3.0 |
| SAP Date: | 21/12/2020 |

### **Notice of Confidential and Proprietary Information:**

The information contained in this document is the property of MEDSENIC. The disclosure of the information to others without written prior approval from MEDSENIC is forbidden.




# STATISTICAL ANALYSIS PLAN DOCUMENT HISTORY

| Version | Date | Author |
|----------|------------|------------------------|
| Final v1 | 13/06/2018 | Myriam Labopin |
| Final v2 | 08/08/2019 | Maëva Dupuis-Deniaud |
| Final v3 | 21/12/2020 | Marine Ragot-Benseghir |




# 1. SIGNATURE PAGE AND APPROVALS

| Written by Marine RAGOT-BENSEGHIR Statistical project leader SOLADIS | Date |
|---|---|
| Approved by Maëva DUPUIS-DENIAUD Biostatistician consultant MDSTAT | Date |
| Sponsor's representative Pr François RIEGER CEO – Scientific Director MEDSENIC | Date |
| Sponsor's representative Dominique GAIDA Clinical Project Manager MEDSENIC | Date |




# 2. SYNOPSIS

| | MEDSENIC |
|---|---|
| | MESSELLIS |
| Sponsor: | 204, avenue de Colmar |
| | F-67100 - Strasbourg |
| | · · |
| Title | Phase II study of first line treatment of Chronic Graft versus Host Disease with Arsenic Trioxide (GvHD-ATO Study) |
| <b>Eudract Number</b> | 2016-002358-18 |
| | Pr Mohamad MOHTY |
| Coordinating investigator | Centre Hospitalier Saint Antoine (AP-HP) |
| | Service d'Hématologie Clinique |
| Phase of development | Phase II |
| | Main Objective |
| | To improve the response rate (complete and partial remission) at 6 months after diagnosis of chronic graft versus host disease (GvHD) and treatment with arsenic trioxide (ATO) in combination with prednisone with or without cyclosporine as a first line treatment |
| | Secondary Objectives |
| Objectives | To evaluate failure-free survival (FFS), defined as death, recurrent or progressive malignancy, or initiation of a new systemic treatment for chronic GvHD |
| | To decrease non-relapse mortality (NRM) of infectious and non-infectious origin |
| | To improve overall survival (OS) and progression-free survival (PFS) |
| | To spare patients from long-term use of corticosteroids (and their long-term side effects) |




| | <ul> <li>To improve quality of life self-reported by patient using the Lee Symptom Scale (LSS) and Functional Assessment of Chronic Illness Therapy with Bone Marrow Transplantation subscale (FACT-BMT)</li> <li>To evaluate tolerability and safety of ATO in combination with prednisone, with or without cyclosporine, in patients with chronic GvHD after allo-SCT</li> </ul> |
|---|---|
| Study design | Prospective, national, multicentre, non-randomized |
| Number of patients planned | 24 patients planned to be included in the study |
| Study centres | 11 sites planned to participate to the study |
| Studied | Inclusion criteria - Adult patients (≥18 years) who have received a first allogeneic stem cell transplantation for a hematological disease (any source of hematopoietic stem cells is authorized; any category of conditioning regimen prior to allo-SCT is authorized; any type of stem cell donors is authorized) - Confirmed diagnosis of first episode of chronic GvHD requiring systemic immunosuppressive therapy (any prior GvHD prophylaxis previously used is accepted). Chronic GvHD diagnosis is defined according to the National Institutes of Health (NIH) Working Group Consensus. |
| population | a/ Performance status evaluation b/ Cutaneous evaluation measured by the percentage of extension or the presence of sclerotic features. If relevant, confirmation with a biopsy should be performed whenever possible c/ Oral symptoms d/ Ocular symptoms e/ Gastro-intestinal symptoms f/ Evaluation of liver involvement manifestations (total bilirubin, transaminases and alkalines phosphatases) g/ Pulmonary function evaluation |




h/ Evaluation of the musculoskeletal manifestations, especially the amplitude of relevant articulations

i/ Genital tract symptoms

- Signed informed consent
- Absence of contra-indications to the use of ATO
- Subjects affiliated with an appropriate social security system
- Men must use a medically acceptable method of contraception throughout the treatment period and for at least 4 months and 10 days following the last treatment administration
- Women who are of childbearing potential must have a negative serum pregnancy test and agree to use a medically acceptable method of contraception throughout the study and for 3 months following the end of the study
- Patient not participating or not having participated in a clinical study in the 30 days prior to his/her inclusion in the study

#### **Exclusion criteria**

- Patient developing acute GvHD (whether early or "late onset" form)
- Patients developing overlap GvHD as defined by the 2015 NIH Working Group Consensus (presence of one or more acute GvHD manifestation in a patient with a diagnosis of chronic GvHD)
- A "mild" form of chronic GvHD not requiring systemic immunosuppressive therapy
- A "moderate" form of chronic GvHD limited to one organ site not requiring systemic immunosuppressive therapy
- Patient receiving mycophenolate mofetil
- Second allogeneic stem cell transplant
- Severe cardiac diseases (congestive heart failure (NYHA class III), recent myocardial infarction (in the past 6 months before the inclusion), histories of unexplained syncope, ...)
- Significant arrhythmias, EKG abnormalities
  - Congenital QT syndromes
  - History or presence of significant ventricular or atrial tachyarrhythmia




| <ul> <li>Clinically</li> </ul> | significant | resting | bradycardia | (<50 | beats | per |
|---|---|---|---|---|---|---|
| minutes) | | | | | | |

- QTc > 450 msec for men and > 470 msec for women on screening EKG
- Right bundle branch block plus left anterior hemiblock, bifascicular block
- Central or peripheral neuropathy
- Neutrophils < 0.5 × 109/L
- Platelets < 50 × 109/L
- Potassium ≤ 4 mEq/l\*
- Magnesium ≤ 1.8 mg/dl\*
- Calcium ≤ 2.15 mmol/l\*
- Hepatic impairment due to a suspected or proven liver damage, other than direct hepatic cGvHD involvement
- PT < 50%
- Renal impairment (creatinine ≥ 100 µmol/l)
- Uncontrolled systemic infection which in the opinion of the investigator is associated with an increased risk of the patients death within 1 month after the start of therapy
- Severe neurological or psychiatric disorders
- Denied informed consent
- Pregnancy
- Women breastfeeding at selection and throughout the treatment period
- \* If abnormal at selection, to be corrected and re-validated following electrolytes infusion, before inclusion and each drug perfusion.

# Investigational product

Arsenic trioxide 10 mg, concentrate for solution for infusion 1 mg/mL (aqueous sterile, clear, colorless).




Arsenic trioxide is administrated either via the marketed product named TRISENOX® or the investigational medicinal product named ARSCIMED®.

Patients under TRISENOX® treatment will not switch to ARSCIMED® treatment nor vice versa:

- Patients already recruited and receiving TRISENOX® will continue receiving only TRISENOX®.
- All patients recruited after this amendment has been approved will receive ARSCIMED<sup>®</sup> only and not TRISENOX<sup>®</sup>.

#### Treatment scheme

As soon as the diagnosis of chronic GvHD requiring systemic immunosuppressive therapy is confirmed, patients will receive in addition to corticosteroids (prednisone) 1/mg/kg/day, with or without cyclosporine A, a daily infusion of ATO 0.15 mg/kg/day on days 1 to 5 (first week), 3 times per week during the second week (for example, days 8, 10 and 12), 2 times per week during the third week (for example, days 15 and 17) and one time during the fourth week (for example, day 24) (the latter four weeks represent one cycle).

ATO should be administered within 10 days of starting prednisone at 1mg/kg/day for cGvHD treatment. Follow-up dates for response assessment and laboratory tests relate to the date of ATO infusion.

Patients who are in partial response after the 1<sup>st</sup> cycle of ATO will be eligible to receive a second cycle of ATO infusions during 4 weeks (similar schedule to first cycle starting around day 60). In another word, a delay of 8 weeks to a maximum of 11 weeks (from the first infusion of ATO) will be observed between the two cycles of ATO therapy.

Response definition is as follows:

- Complete remission (CR) is defined as complete disappearance of any sign of chronic GvHD
- Partial remission (PR) is defined as improvement of 1 or more point on a 4 to 7-point scale or improvement of 2 or more points on a 10 to 12-points scale in at least 1 organ or site without progression in any other organ or site. For patients with Bronchiolitis Obliterans Syndrome (BOS), an absolute




improvement in % FEV1 of 10% predicted or more (eg, 50% to 60%) is considered a PR as long as the initial % FEV1 is < 70%. Normalization (≥ 80%) is considered a CR.

- Failure is defined as death, recurrent or progressive malignancy or the irritation of new systemic treatment for chronic GvHD. Increased dosing of existing treatment will not be considered as failure. Early failure is defined as failure within 2 weeks after the end of the first ATO cycle.

Indications for secondary systemic treatment of chronic GvHD

Secondary systemic immunosuppressive treatment or other systemic treatment for control of chronic GvHD will be given at the discretion of the investigator in consultation with the GvHD team. In general, secondary systemic treatment is not indicated as long as there is continuing improvement in at least one manifestation of chronic GvHD and no progression of any other manifestations.

#### Primary endpoint

 Evaluation of response rate (complete and partial remission) of chronic GvHD at 6 months after diagnosis of chronic GvHD and treatment with arsenic trioxide (ATO) in combination with prednisone, with or without cyclosporine, as first line treatment.

#### Secondary endpoints

#### Study endpoints

- Percentage of patients with documented failure free survival (FFS), defined as death, recurrent or progressive malignancy, or the initiation of a new systemic treatment for chronic GvHD
- Corticosteroids dosage and percentage of reduction in corticosteroids dosage at 6 and 12 months after diagnosis of chronic GvHD and treatment with ATO as first line treatment
- Cumulative dosage and percentage of reduction in corticosteroids dosage at 6 and 12 months after diagnosis of chronic GvHD and treatment with ATO as first line treatment
- OS and PFS at 6 and 12 months after diagnosis of chronic GvHD and treatment ATO as first line treatment




| - | Descriptive | analysi | s of q | uality of life | para | meters | s at | inclus | sion, |
|---|---|---|---|---|---|---|---|---|---|
| | at 6 and 14 | weeks, | and a | at 6, 9 and 1 | 12 mo | nths a | fter | diagn | osis |
| | of chronic | GvHD | and | treatment | with | ATO | as | first | line |
| | treatment. | | | | | | | | |

 Tolerability and safety of ATO in combination with prednisone, with or without cyclosporine, in patients with chronic GvHD after allo-SCT.

#### Sample size calculation

Based on results from the literature, the hypothesis for the primary endpoint is an improvement in response rate (complete an partial remission) at 6 months after the diagnosis of chronic GvHD and start of corticosteroids, ATO, with or without cyclosporine, from 60% to 85%. Using a one step A Hern procedure (and anticipating a dropout rate around 10%), 24 (21+3) patients are needed (A'Hern RP, 2001).

If the number of successful cases is 17 or more among the 21 patients, the hypothesis that the CR rate at 6 months is less than 60% is rejected with a target error rate of 0.05 (alpha probability). The beta probability in this case is 0.2.

#### Statistical analyses

# Statistical methods

Every patient included in the study and who has received at least one infusion of ATO will be taken into account at time of data analysis. A descriptive analysis will be conducted on the following parameters:

- Patients and transplant characteristics
- Primary and secondary endpoints

Patients who do not receive any injection of ATO will not be analysed and will be replaced to obtain 24 patients provided in the statistical analysis.

Qualitative data will be described in frequency and percentage and will be represented using histograms or diagrams of distribution. Quantitative data will be described using the calculations of average, standard deviation, median, and extreme values.

The toxicities rate will be calculated and will be given with their 95% confidence intervals.




| The probabilities of survival will be estimated by the Kaplan-Meier method and by calculating the cumulative incidences for relapse/progression, and non-relapse mortality incidence. |
|---|
| The total duration of the study is expected to be 46 months (duration of recruitment: 34 months and study duration for a considered patient: 12 months) |
| First patient first visit: September 2016 |
| Last patient last visit: June 2020 |
| Database lock: December 2020 |
| Clinical study Report: March 2020 |




# 3. TABLE OF CONTENTS

| 1. | SIGNATURE PAGE AND APPROVALS | 4 |
|------------|--------------------------------------------------|----|
| 2. | SYNOPSIS | 5 |
| 3. | TABLE OF CONTENTS | 13 |
| 4. | LIST OF ABBREVIATIONS AND DEFINITION OF TERMS | 16 |
| 5. | ETHICS | 17 |
| 5.1 | REGULATORY AUTHORITIES APPROVAL (CPP AND ANSM) | 17 |
| 5.2 | INFORMED CONSENT | 18 |
| 5.3 | INVESTIGATORS RESPONSABILITIES | 18 |
| 5.4 | SPONSOR RESPONSABILITIES | 20 |
| 5.5 | BIOCOLLECTIONS | 20 |
| 5.6 | ARCHIVING | 20 |
| 6. | INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE | 21 |
| 7. | INTRODUCTION | 22 |
| 8. | STUDY OBJECTIVES AND ENDPOINTS | 24 |
| _ | OBJECTIVES | 24 |
| 8 | .1.2 Secondary objectives | 24 |
| <b>8.2</b> | ENDPOINTS | |
| | 2.2 Secondary endpoints | 25 |




| 9. INVESTI | GATIONAL PLAN | . 27 |
|---|---|---|
| 9.1 OVERA | LL STUDY DESIGN AND PLAN | 27 |
| 9.2.1 Inclus | TION OF STUDY POPULATIONsion criteriasion criteria | 28 |
| 9.3 TREATI | MENTS | 30 |
| 9.3.2 Identi | ments administeredity of Investigational Product(s) | 32 |
| 9.3.4 Metho | nistrationod of Assigning Patients to Treatments Groupsing | 33 |
| | and Concomitant Therapy | |
| | CY AND SAFETY VARIABLESacy and Safety Measurements Assessed and Schedule of Assessments | |
| 9.5 DATA C | QUALITY ASSURANCE | 40 |
| 9.5.2 AUDI<br>9.5.3 MON | CLINICAL PRACTICETINGITORING | 40<br>40 |
| 12.4 STATIS | TICAL ANALYSIS METHODES PLANNED IN THE PROTOCOL AND ON OF SAMPLE SIZE | 43 |
| 12.5 CHANG | ES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSIS | 45 |
| 10. PATIENT | rs | . 46 |
| 10.1 DISPOS | SITION OF PATIENTS | 46 |
| 10.2 PROTO | COL DEVIATIONS | 47 |
| 11. EFFICAC | CY EVALUATION | . 48 |
| 11.1 ANALY | SES POPULATIONS | 48 |
| 11.2.1 De<br>11.2.2 Ba | BRAPHIC AND OTHER BASELINE CHARACTERISTICS | 49<br>50 |




| 11.3 | ATO AND ASSOCIATED TREATMENTS | 61 |
|---|---|---|
| 11 | 1.3.1 Arsenic trioxide therapy | 61 |
| 11 | 1.3.2 Associated treatment | 66 |
| 11.4 | EFFICACY ANALYSIS | 69 |
| | 1.4.1 Primary Endpoint analysis | |
| | 1.4.2 Secondary Endpoint analyses | |
| 12. | SAFETY EVALUATION | 95 |
| 12.1 | ADVERSE EVENTS | 95 |
| 12.2 | LABORATORY PARAMETERS | 97 |
| 12.3 | PHYSICAL EXAMINATION | 99 |
| 13. | DISCUSSION AND OVERALL CONCLUSIONS | 101 |
| 14. | TABLES, FIGURES AND GRAPHS | 102 |
| 14.<br>14.1 | | |
| | TABLES | 102 |
| 14.1<br>14.2 | TABLES | 102<br>105 |
| 14.1<br>14.2<br>15. | TABLESFIGURES AND GRAPHS | 102<br>105 |
| 14.1<br>14.2<br>15.<br>16. | TABLES FIGURES AND GRAPHS REFERENCE LIST | 102<br>105<br>109 |
| 14.1<br>14.2<br>15.<br>16. | TABLES FIGURES AND GRAPHS REFERENCE LIST LISTINGS | 102<br>105<br>109<br>110 |
| 14.1<br>14.2<br>15.<br>16. | TABLES | 102105109110111 |
| 14.1<br>14.2<br>15.<br>16.<br>17.<br>17.1 | TABLES | 102105110110111 |
| 14.1<br>14.2<br>15.<br>16.<br>17.<br>17.1 | TABLES | 102105109110111111 |




#### 4. LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

AE Adverse Event

ALAT/SGPT Alanine Amino-Transferase

Allo-SCT Allogeneic Stem-Cell Transplantation
APL Acute Promyelocytic Leukemia
ASAT/SGOT Aspartate Amino-Transferase

ATO Arsenic Trioxide

ATRA All-trans Retinoic Acid (tretinoin)

CBC Complete Blood Count

cGvHD Chronic Graft Versus Host Disease

CMV Cytomegalovirus CR Complete Remission

DLI Donor Lymphocytes Infusion

EBV Epstein Barr Virus

e-CRF Electronic Case Report Form

EKG Electrocardiogram

FACT-BMT Functional Assessment of Chronic Illness

Therapy with Bone Marrow Transplantation

subscale

FAS Full Analysis Set

FEV Forced Expiratory Volume
FFS Failure-free Survival
GHVD Graft Versus Host Disease

Hep Hepatitis

HLA Human Leucocyte Antigen HY Y-chromosome—encoded

ICH International Conference on Harmonization

IQR inter-quartile range

IVIG Intravenous Immunoglobulin

HSCT Hematopoietic Stem Cell Transplantation

LSS Lee Symptom Scale

MedDRA Medical Dictionary for Regulatory Activities

NIH National Institutes of Health
NRM Non-relapse Mortality
OS Overall Survival

PDC Plasmacytoid Dendritic Cells
PFS Progression-free Survival
PI Principal Investigator

PP Per Protocol
PR Partial Remission

RIC
Reduced Intensity Conditioning
ROS
Reactive Oxygen Species
SAE
Serious Adverse Event
TRM
Transplant-related Mortality
WHO
World Health Organization




#### 5. ETHICS

The study will be conducted according to the European Union directive (ICH Harmonized Tripartite Guideline for Good Clinical Practice, (17.01.1997)). The study has to be conducted in compliance with the protocol, GCP and all applicable regulatory requirements:

- Helsinki declaration from 1964, revised in Washington in 2002,
- GCP of the International Harmonization Conference (ICH E6, 17/07/96),
- European Directive (2001/20/CE) on the conduct of clinical trials,
- French law n° 2004-801 dated 6 August 2004,
- French bioethics law no 2004-800 dated 6 August 2004.

Accordingly, investigating physicians have to provide direct access to study documents to monitoring, audits, institutional internal control, external authorities, and the members of the ethical committee. Written informed consent by the patient is mandatory.

The coordinating investigator and all investigators will be given an up-to-date investigator's brochure containing full details of the status of the pre-clinical and clinical knowledge of the study medication. As soon as new information is obtained, an updated version will be supplied or an amendment added to the existing investigator's brochure.

## 5.1 REGULATORY AUTHORITIES APPROVAL (CPP AND ANSM)

No patient may be included in the study before the respective requirements of the national health authorities are fulfilled. The study will begin only after the positive vote of the responsible Ethics Committee (CPP) and after the approval by the appropriate national health authority (ANSM).

The protocol has to be followed strictly, protocol violations have to be documented and the reason has to be given (e.g. emergency measures). Any changes in the protocol can only be performed by the principle investigator or the protocol writing committee. Any




subsequent changes will be reported or submitted for approval to the ethical committee and to local and national authorities.

#### 5.2 INFORMED CONSENT

Written informed consent is obtained by each patient before inclusion into the study. Using patient information sheets, as well as personal oral explanation by a local investigator at the patient's transplant centre, the patient will be informed of the aims and the investigational nature of the study, the exact procedures that will be done during treatment and evaluation, the possible risks and side effects, and of alternative treatment options. They will be informed as to the strict confidentiality of their patient data, but that authorized individuals other than their treating physician may review their medical records for study purposes. Further, the patient will be informed that their anonymized data will be scientifically analyzed and published. It will be emphasized that the participation is voluntary and that consent can be withdrawn by the patient at any time without explanation of the reason. The patient is allowed to refuse further participation in the protocol, whenever he/she wants. The patient's further treatment will not be influenced by this decision.

#### 5.3 INVESTIGATORS RESPONSABILITIES

In collaboration and according to the Standard Operating Procedure (SOP) of the sponsor, a detailed list of delegation of responsibilities has been established. It is held by the sponsor, who is finally responsible for the correct performance of delegated responsibilities by the respective persons or institutions. A copy of this list will be delivered to the participating institutions.

The investigator of each institution undertakes to conduct the study according to the protocol which was approved by the ethics (CCP) and health authorities (ANSM). The




investigator must not make any changes to the protocol without the permission of the sponsor and without the CCP has given a favorable opinion on the proposed amendments.

It is the responsibility of the investigator responsible for the study in the participating centre:

- To provide his curriculum vitae as well as co-investigators
- To identify team members, who will participate in the study and define their responsibilities
- To start recruiting patients after authorization of the sponsor
- To try to include the required number of patients within the period of recruitment

It is the responsibility of each investigator:

- To obtain the informed consent dated and signed personally by the patient before any selection process specific to the study
- To fill in an electronic case report form (e-CRF) for each patient included in the study and allow direct access to source documents to validate e-CRF data \_ To correct, sign and date the correction(s) of the e-CRF for each patient enrolled
- To notify the sponsor of any SAE(s) within the time required
- To accept regular monitoring visits and possibly those of auditors mandated by the sponsor or inspectors from authorities

All documentation on the study (protocol, consents, notebooks observation, file investigator, etc.) and original documents (laboratory results, x-rays, minutes of consultations, review reports...) must be kept in a safe place and considered confidential material.

The Investigator will maintain the confidentiality of the identity of subjects enrolled in the study and the information contained in the study records.




#### 5.4 SPONSOR RESPONSABILITIES

It is the responsibility of the sponsor to:

- Subscribe insurance to cover its liability for the harmful consequences of research
- Provide the investigators with all information necessary to conduct the research
- Apply for authorization from a relevant CPP
- Apply for authorization from ANSM
- Inform the Directors and Pharmacists of health facilities
- Inform ANSM of any serious incidents that may be due to research

#### 5.5 BIOCOLLECTIONS

Biological samples collected for the immunological assessment will be stored in a biocollection. The patient informed consent will be collected and the samples will be stored in one of the biocollections of Assistance Publique-Hôpitaux de Paris: the Hematology biobank approved by INCa and located at the Saint-Antoine Hospital (Declaration N  $^{\circ}$  DC-2009-963 and authorization N  $^{\circ}$  AC-2013-1992).

The Sponsor shall finance the study and endorses a policy of insurance covering the financial consequences of its civil liability in accordance with regulations in order to guarantee against possible damage resulting from the research.

Non-compliance with the Research Legal Conditions is a cause for guarantee exclusion.

#### 5.6 ARCHIVING

The data archiving will be under the responsibility of the investigator and, as required by law.

Data will be kept for a minimum of 15 years after the end of the study.




# 6. INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE

| Sponsor | MEDSENIC |
|---------------------------------|--------------------------------|
| | 204, avenue de Colmar |
| | F-67100 Strasbourg |
| | Tel: + 33 (0) 1 79 25 14 42 |
| CEO- Scientific Director | Pr François Rieger |
| | Mail: |
| Executive Director | Véronique Pomi |
| | Mail: |
| Clinical Project Leader | Dominique Gaïda, PhD |
| | Mail: |
| Coordinating Investigator | Pr Mohamad MOHTY |
| | Service d'Hématologie Clinique |
| | Hôpital Saint Antoine AP-HP |
| | F-75012 – Paris |
| | Tel: |
| Contract Reasearch Organization | PopsiCube – Fovea |
| | 6 rue Jean-Pierre Timbaud |
| | Le Campus – Bât A1 Sud |
| | F-78180 Montigny le Bretonneux |
| | Tel: |
| | Fax: |




#### 7. INTRODUCTION

Chronic Graft-versus-Host Disease (GvHD) is one of the most common and clinically significant complication affecting long-term survivors of allogeneic stem cell transplantation (allo-SCT). Chronic GvHD (cGvHD) is the cause of death in up to one third of all long-term survivors after transplantation for leukemia and is consistently associated with decreased quality of life, impaired functional status, ongoing need for immunosuppressive medications and infectious complications. Standard first line systemic treatment for cGvHD is orally administered corticosteroids (prednisolone 1 mg/Kg/d) and cyclosporine, with a median duration reported between 18 and 23 months. Therapy with corticosteroids is often unrewarding and the toxicities from prolonged corticosteroid administration are great. Chronic GvHD emerges from alloreactive processes between donor-derived immune cells and host cell populations. While its pathophysiology is still poorly understood, data in humans support a role of both T and B cells in a highly complex network. How these T- and B-cell networks interact has not been resolved.

Arsenic derivatives have been identified as compounds with therapeutic potential for over 2000 years in Greek and Chinese medicine. The combination of ATO and oral all-trans retinoic acid tretinoin [ATRA]) currently constitutes the standard of care for most patients with newly diagnosed and/or relapsed acute promyelocytic leukemia (APL). The use of ATO has also been explored in many other hematologic malignancies and in solid tumors. Its role has also been explored in murine models of autoimmune and autoinflammatory diseases. Chronic GvHD presents clinical features that mimic autoimmune diseases such as systemic sclerosis, lupus erythematosus or Sjögren syndrome, and autoimmune-like manifestations are a defining characteristic of cGvHD. In a murine model of chronic GvHD, ATO effect was mediated through the depletion of glutathione and the overproduction of H2O2 that killed activated CD4+ T cells, in particular Th17 cells, and PDC, two key cells in chronic GvHD pathophysiology initiation. Furthermore, autoantibody production was also inhibited by ATO in this model, suggesting that ATO also triggers B cells death in a phenomenon which cooperates for controlling chronic GvHD.




This leads to the hypothesis that ATO delivered during the course of the disease or even early at diagnosis of chronic GvHD- and possibly in prevention of cGvHD before its detection- will be an effective treatment. To test this hypothesis, we proposed this study of ATO in combination with corticosteroids as first line therapy for newly diagnosed chronic GvHD after allo-SCT. We hypothesized that the addition of ATO to prednisone for the initial treatment of chronic GvHD will increase the overall response rate and enable a more rapid and effective corticosteroids taper. We authorized the use of cyclosporine A, as a somewhat widely adopted measure, due to its use for its supposed possible beneficial action on acute GvHD in the early weeks after allografting and sometimes continuously maintained in spite of recognized inefficacy to influence the course of the autoimmune processes going on under the designation of cGvHD.




#### 8. STUDY OBJECTIVES AND ENDPOINTS

#### 8.1 OBJECTIVES

#### 8.1.1 Primary objective

The primary objective is to improve the response rate (complete and partial remission) at 6 months after diagnosis of chronic GvHD and treatment with arsenic trioxide (ATO) in combination with prednisone with or without Ciclosporin as first line treatment.

The aim of this study is to assess whether ATO allows improving response rate at 6 months after the diagnosis of chronic GVHD from 60% (historical rate) to 85%.

#### 8.1.2 Secondary objectives

The secondary objectives are:

- To evaluate failure-free survival (FFS), defined as death, recurrent or progressive malignancy, or initiation of a new systemic treatment for chronic GvHD
- To decrease non-relapse mortality (NRM) of infectious and non-infectious origin
- To improve overall survival (OS) and progression-free survival (PFS)
- To spare patients from long-term use of corticosteroids (and their long-term side effects)
- To improve quality of life self-reported by patient using the Lee Symptom Scale (LSS) and Functional Assessment of Chronic Illness Therapy with Bone Marrow Transplantation subscale (FACT-BMT)
- To evaluate tolerability and safety of ATO in combination with prednisone, with or without Ciclosporin, in patients with chronic GvHD after allo-SCT.

#### 8.2 ENDPOINTS

#### 8.2.1 Primary endpoint

The primary endpoint is the evaluation of response rate (CR and PR) at 6 months after the first ATO infusion, with no secondary systemic therapy at any time before M6.

NIH grade of chronic GVHD will be used for the exact definition of this endpoint.




- Complete remission (CR) is defined as complete disappearance of any sign of chronic GvHD
- Partial remission (PR) is defined as improvement of 1 or more point on a 4 to 7points scale or an improvement of 2 or more points on a 10 to 12-points scale in at
  least 1 organ or site without progression in any other organ or site.
- More details for response determination are given in the following table:

| Organ | Complete Response | Partial Response | Progression |
|---|---|---|---|
| Skin | NIH Skin Score 0 after | Decrease in NIH Skin Score | Increase in NIH Skin Score by 1 or |
| | previous involvement | by 1 or more points | more points, except 0 to 1 |
| Eyes | NIH Eye Score 0 after | Decrease in NIH Eye Score | Increase in NIH Eye Score by 1 or |
| | previous involvement | by 1 or more points | more points, except 0 to 1 |
| Mouth | NIH Modified OMRS 0 after | Decrease in NIH Modified OMRS | Increase in NIH Modified OMRS |
| | previous involvement | of 2 or more points | of 2 or more points |
| Esophagus | NIH Esophagus Score 0 after | Decrease in NIH Esophagus | Increase in NIH Esophagus Score |
| | previous involvement | Score by 1 or more points | by 1 or more points, except 0 to 1 |
| Upper GI | NIH Upper GI Score 0 after | Decrease in NIH Upper GI | Increase in NIH Upper GI Score |
| | previous involvement | Score by 1 or more points | by 1 or more points, except 0 to 1 |
| Lower GI | NIH Lower GI Score 0 after | Decrease in NIH Lower GI | Increase in NIH Lower GI Score by 1 |
| | previous involvement | Score by 1 or more points | or more points, except from 0 to 1 |
| Liver | Normal ALT, alkaline | Decrease by 50% | Increase by 2 × ULN |
| | phosphatase, and Total | | |
| | bilirubin after previous | | |
| | elevation of 1 or more | | |
| Lungs | - Normal %FEV1 after | - Increase by 10% predicted | - Decrease by 10% predicted |
| Lungs | previous involvement | absolute value of %FEV1 | absolute value of %FEV1 |
| | - If PFTs not available, NIH | - If PFTs not available, decrease | - If PFTs not available, increase in |
| | Lung Symptom Score 0 | in NIH Lung Symptom Score | NIH Lung Symptom Score by 1 |
| | after previous involvement | by 1 or more points | or more points, except 0 to 1 |
| Joints and fascia | Both NIH Joint and Fascia | Decrease in NIH Joint and Fascia | Increase in NIH Joint and Fascia |
| | Score 0 and P-ROM score | Score by 1 or more points or | Score by 1 or more points or |
| | 25 after previous involvement | increase in P-ROM score by 1 | decrease in P-ROM score by 1 |
| | by at least 1 measure | point for any site | point for any site |
| Global | Clinician overall severity score 0 | Clinician overall severity score | Clinician overall severity score |
| | continuo oreitan severity sevice o | decreases by 2 or more points | increases by 2 or more points |
| | | on a 0-10 scale | on a 0-10 scale |

ULN indicates upper limit of normal.

### 8.2.2 Secondary endpoints

- OS is defined as the time from first infusion of ATO to death, regardless of the cause
- FFS is defined as related death, progression, or initiation of a new systemic treatment for chronic GvHD
- PFS is defined as survival with no evidence of relapse or progression of the original disease




- Corticosteroids dosage and percentage of reduction in corticosteroids dosage at 6 and 12 months after diagnosis of chronic GvHD and treatment with ATO as first line treatment
- Quality of life parameters using FACT-BMT and Lee Symptom Scale scores at 6 and 14 weeks, 6, 9 and 12 months after first infusion of ATO
- Tolerability and safety of ATO


#### 9. INVESTIGATIONAL PLAN

#### 9.1 OVERALL STUDY DESIGN AND PLAN

The study GMED16-001 is a prospective, national, multicenter, non-randomized phase II study that will include a total number of 24 patients.

The duration of participation panned is as follows:

- Duration of recruitment: 34 months
- Study duration for a considered patient: 12 months
- Total duration of the study: 46 months

Several visits are scheduled in the study as follows:

- At the time of diagnosis for the screening visit
- Follow-up visits to be performed every week during ATO treatment
- Follow-up visits to be performed every 2 weeks from second to third month of ATO treatment
- Follow-up visits to be performed every month from the fourth to sixth month of ATO treatment
- Follow-up visits to be performed every 3 months: at 9 months and 12 months (final visit)






Arsenic trioxide is administrated either via the marketed product named TRISENOX® or the investigational medicinal product named ARSCIMED®.

#### 9.2 SELECTION OF STUDY POPULATION

#### 9.2.1 Inclusion criteria

Patients will be eligible for inclusion in this study if the patient met all the following criteria:

- Adult patients (≥18 years) who have received a first allogeneic stem cell transplantation for a hematological disease (any source of hematopoietic stem cells is authorized; any category of conditioning regimen prior to allo-SCT is authorized; any type of stem cell donors is authorized)
- Confirmed diagnosis of first episode of chronic GvHD requiring systemic immunosuppressive therapy (any prior GvHD prophylaxis previously used is accepted). Chronic GvHD diagnosis is defined according to the National Institutes of Health (NIH) Working Group Consensus.
- Signed informed consent
- Absence of contra-indications to the use of ATO
- Subjects affiliated with an appropriate social security system
- Men must use a medically acceptable method of contraception throughout the treatment period and for at least 4 months and 10 days following the last treatment administration
- Women who are of childbearing potential must have a negative serum pregnancy test and agree to use a medically acceptable method of contraception throughout the study and for 3 months following the end of the study
- Patient not participating or not having participated in a clinical study in the 30 days prior to his/her inclusion in the study

#### 9.2.2 Exclusion criteria

Patients fulfilling ONE or MORE of the following criteria will not be included in the study:

• Patient developing acute GvHD (whether early or "late onset" form)




- Patients developing overlap GvHD as defined by the 2015 NIH Working Group Consensus (presence of one or more acute GvHD manifestation in a patient with a diagnosis of chronic GvHD)
- A "mild" form of chronic GvHD not requiring systemic immunosuppressive therapy
- A "moderate" form of chronic GvHD limited to one organ site not requiring systemic immunosuppressive therapy
- Patient receiving mycophenolate mofetil
- Second allogeneic stem cell transplant
- Severe cardiac diseases (congestive heart failure (NYHA class III), recent myocardial infarction (in the past 6 months before the inclusion), histories of unexplained syncope, ...)
- Significant arrhythmias, EKG abnormalities
  - Congenital QT syndromes
  - History or presence of significant ventricular or atrial tachyarrhythmia
  - Clinically significant resting bradycardia (<50 beats per minutes)
  - QTc > 450 msec for men and > 470 msec for women on screening EKG
  - Right bundle branch block plus left anterior hemiblock, bifascicular block
- Central or peripheral neuropathy
- Neutrophils < 0.5 × 109/L</li>
- Platelets < 50 × 109/L</li>
- Potassium ≤ 4 mEq/l
- Magnesium ≤ 1.8 mg/dl
- Calcium ≤ 2.15 mmol/l
- Hepatic impairment due to a suspected or proven liver damage, other than direct hepatic cGvHD involvement
- PT < 50%</li>
- Renal impairment (creatinine ≥ 100 µmol/l)
- Uncontrolled systemic infection which in the opinion of the investigator is associated with an increased risk of the patients death within 1 month after the start of therapy
- Severe neurological or psychiatric disorders




- Denied informed consent
- Pregnancy
- Women breastfeeding at selection and throughout the treatment period

#### 9.3 TREATMENTS

#### 9.3.1 Treatments administered

Arsenic trioxide (ATO) is administrated either via a marketed product, i.e. TRISENOX®, or an Investigational Medicinal Product, i.e. ARSCIMED®.

TRISENOX® was administered to patients from the start of the clinical trial. ARSCIMED® will be administered to patients included in the clinical trial after approval from the ANSM for its use in this clinical trial. Patients under TRISENOX® treatment will not switch to ARSCIMED® treatment nor vice versa.

- All patients already included in the trial and who received TRISENOX® will continue with TRISENOX® until completion of their participation in the clinical trial.
- All patients recruited after this amendment has been approved will receive ARSCIMED® only and not TRISENOX®.

TRISENOX® and ARSCIMED® have the same active substance, excipients, dosage form and route of administration (Summary of Product Characteristics (Trisenox)) and Investigator brochure (ARSCIMED®) for details) and are considered equivalent. The decision in switching to ARSCIMED® during the clinical trial is based on the fact that the availability of ARSCIMED®, treatment being developed by MEDSENIC in the population included in this trial, will avoid repeated and further impact on recruitment in the study related to any further supply disruptions of TRISENOX®, as it occurred in 2014 and again in 2017.




Both formulations (TRISENOX® and ARSCIMED® are adjusted to pH 8 with dilute hydrochloric acid. Whereas TRISENOX® is manufactured by TEVA and supplied as a glass ampoule; ARSCIMED® is manufactured by IRPF¹-Toulouse and supplied as a glass vial. Further information on ARSCIMED® is available in the Investigational Medical Product Dossier of this product.




### 9.3.2 Identity of Investigational Product(s)

The investigational medication has the following characteristics:

- ATC code: LOIXX27
- Pharmacotherapeutic group: other antineoplastic agents
- Form/Presentation: concentrate for solution for intravenous infusion / 1 mg/1 mL / 10 mL
- Excipients: sodium hydroxide, hydrochloric acid as pH adjuster and water for injections

#### 9.3.3 Administration

- 0, 15 mg/kg/infusion on days I to 5 (first week), 3 times per week during the second week (for example, days 8, 10 and 12), 2 times per week during the third week (for example, days 15 and 17) and one time during the fourth week (for example, day 24), in addition to Ciclosporin A (if relevant) and corticosteroids. The latter four weeks represent one cycle of 11 administrations.
- Must be administered intravenously over 1-2 hours. The infusion duration may be extended up to 4 hours if vasomotor reactions are observed. A central venous catheter is not required. Patients must be hospitalized at the beginning of treatment due to ensure adequate monitoring.
- Aseptic technique must be strictly observed throughout handling of ATO since no preservative is present.
- Must be diluted with 100 to 250 mL of glucose 50 mg/mL (5%) solution for injection or sodium chloride 9 mg/mL (0.9%) solution for injection immediately after withdrawal from the ampoule for single use only. Unused




portions of each ampoule must be discarded properly. Unused portions for later administration must not be saved.

- Must not be mixed with or concomitantly administered in the same intravenous line with other medicinal products.
- The diluted solution must be clear and colorless. All parenteral solutions
  must be inspected visually for particulate matter and discoloration prior to
  administration. The preparation must not be used if foreign particulate matter
  is present.
- Should be administered within 10 days of starting prednisone at I mg/kg/day for cGvHD treatment. Treatment with persistent prednisone (or equivalent) at doses lower than 1 mg/kg/day at the time of enrollment is allowed (i.e patient was treated for acute GvHD with prednisone and developed evolving chronic GvHD).
- A delay of 8 weeks to a maximum of 1 1 weeks (from the first infusion of ATO) will be observed between the two cycles of ATO therapy.

# 9.3.4 Method of Assigning Patients to Treatments Groups

Not Applicable

9.3.5 Blinding

Not Applicable




### 9.3.6 Prior and Concomitant Therapy

#### 9.3.6.1 Ciclosporin A

- Ciclosporin A will be delivered using local standard criteria, (if relevant).
  However:
  - Ciclosporin level should lie within the therapeutic range (i.e. 200-400 ng/mL): to harmonize CSA target levels
  - Ciclosporin-induced renal insufficiency should lead to dose adjustment and even temporary withdrawal of the drug
- Suggested guidelines for initial dose of Ciclosporin A:

Oral administration of Ciclosporin should continue for patients who are being treated with Ciclosporin at the time of enrolment, or if it is relevant. the administration should commence initially at 6mg/kg daily.

- Monitoring of Ciclosporin level:
  - Concentrations of Ciclosporin in the plasma may be monitored at the discretion of the investigator. Dose adjustments may be made to maintain Ciclosporin concentrations at 200-400 ng/ml. Monitoring may be especially helpful in patients with renal impairment and in patients being treated with medications that may affect the concentration of Ciclosporin.
  - Medications that could increase the concentration of Ciclosporin include diltiazem, nicardipine, verapamil, metoclopramide, ketoconazole, fluconazole, itraconazole, erythromycin and methylprednisolone.
  - Medications that could decrease the concentration of Ciclosporin include rifampycin, phenytoin, phenobarbital and carbamazepine.
- Deviations from guidelines for administration of Ciclosporin Deviations from the above guidelines may be made at the discretion of the investigator in consultation with the transplant centre. Toxicity associated with the




administration of Ciclosporin may require dose adjustments, which should be managed according to individual transplant centre practice.

#### 9.3.6.2 Prednisone

- ➤ The initial dose of prednisone is 1.0 mg/kg/day, this dose should be maintained for 2 weeks, after which a tapering schedule should commence up until response assessment at 6 weeks, after which treatment is as follows:
- CR: continue tapering of Prednisone dose (see Table below)
- No CR: maintain Prednisone dose at 1 mg/kg/day on alternate days or 0.5 mg/kg/day every day
  - Usual prevention of steroid-induced gastro-intestinal (GI) side effect should be given (omeprazole or other drugs, according to local practice).
- The investigator will determine the regimen for administration of prednisone after enrolment in the study. The following taper schedule is given as a general guideline:

#### **Prednisone Taper Schedule**

| Week | Dose (mg/kg actual body weight/day) |
|---|---|
| 0 | 1.0 qod |
| 2 | 0.75 qod |
| 4 | 0.65 qod |
| 6 | 0.50 qod (if CR, continued tapering of corticosteroids dose) |
| | 0.50 qod (if No CR, maintain this dose until resolution of all reversible clinical manifestations or adjust the required dose) |




| 8 | 0.40 qod |
|----|----------|
| 10 | 0.30 qod |
| 12 | 0.20 qod |
| 14 | 0.15 qod |
| 20 | 0.0 |

- The investigator should examine the patient before each reduction in the dose of prednisone. If there is exacerbation or recurrence of chronic GvHD at any step of the taper, the dose of prednisone should be increased by 2 levels with daily administration for 2-4 weeks, followed by resumption of alternate day administration. Prednisone may be discontinued after 2 weeks of treatment at a dose of 0.15 mg/kg every other day. Qod prednisone dosing is not required, and the use of qod dosing is at the discretion of the investigator. It is suggested, but not required, that patients taper off steroids before tapering of other immunosuppressive medications.
- Toxicity associated with the administration of prednisone should be managed according to individual transplant center practice.

# 9.3.6.3 Preventive treatments for infections

- Antibiotic prophylaxis for prevention of Pneumocystis pneumonia and infections with encapsulated organisms must be given to all patients until 6 months after discontinuation of all systemic immunosuppressive treatment. Suggested antibiotic regimens are: Trimethoprim/Sulfamethoxazole DS I tab PO qMWF, or if sulfa allergic, Atovaquone 1500 mg PO qMWF or Pentamidine 300 mg inhaled q4 weeks. Additional prophylactic antibiotics are at the discretion of the physician.



- Prophylactic antiviral and antifungal medications must also be given until the steroid dose is stable < 0.15 mg/kg/day. All patients who are at risk of CMV infection should be monitored for occult CMV infection, and appropriate treatment should be instituted per institutional practice. Populations at risk of CMV infection include all CMV seropositive patients, all CMV-seronegative patients with CMV-seropositive donors, and all patients receiving blood product transfusions from CMV-seropositive donors.
- Antifungal prophylaxis: No specific antifungal prophylaxis is recommended. In case it is the routine policy of a centre to give an antifungal prophylaxis in patients with chronic GvHD (i.e., fluconazole, oral amphotericin B, itraconazole, posaconazole or other drugs for which there are published data of controlled trials showing the antifungal prophylaxis of this drug in allo-SCT patients), it is required that this policy is being documented in the CRF and the same policy be applied to all the patients included in the centre.
- In all cases, physicians can refer to the recommendations made by the European Conference on Infections in Leukemia (ECIL). The full version is available on the website of the EBMT: https://www.ebmt.org/Contents/Resources/Library/ECIL/Pages/ECIL.aspx
- All treatments given for prevention of infectious complications must be reported in the electronic CRF of the study.

## 9.3.6.4 Prohibited concomitant treatments

- Patient receiving mycophenolate mofetil
- Any other investigational study drugs than ATO




### 9.4 EFFICACY AND SAFETY VARIABLES

# 9.4.1 Efficacy and Safety Measurements Assessed and Schedule of Assessments

Patients will undergo the procedures and examinations which must be performed as shown in the following flow chart:

| | Selection (V1) (10 days before ATO treatment) | During ATO<br>treatment<br>(1st and<br>2nd cycles) | Every 2<br>weeks<br>(from M2<br>to M3)<br>± 5 days | Every<br>month<br>(M4,<br>M5,<br>M6)<br>± 5<br>days | At 6 and<br>14 weeks<br>and every<br>3 months<br>(M6, M9,<br>M12)<br>± 5 days | Study<br>drop-<br>out ± 5<br>days |
|---|---|---|---|---|---|---|
| Information and patient consent | * | | | | | |
| Inclusion/exclusion criteria check | * | | | | | |
| Socio-demographics | * | | | | | |
| Concomitant diseases | * | | _ | | | |
| Recipient, Donor and<br>Transplant characteristics <sup>10</sup> | * | | | | | |
| Diagnosis & Scoring of chronic GvHD | * | | | | | |
| Chronic GvHD activity assessment form A | * | | | | * | * |
| Chronic GvHD activity assessment form B | * | | | | * | * |
| Lee Symptom scale | * | | | | * | * |
| FACT-BMT | * | | | | * | * |
| Physical examination | * | *1 | * | * | * | * |
| EKG – QTc1 measurement | * | *1 | * | | | |
| Hematology3 | * | *9 | * | * | * | * |
| Biochemistry4 | * | *2/9 | * | * | * | * |
| Coagulation test5 | * | *9 | * | * | * | * |
| Infectious disease surveillance | * | *2 | | * | * | * |
| Serum immunoglobulin level | * | | | * | * | * |
| Autoantibodies (AAN, ANCA) | * | *2 | | * | * | * |
| Serum pregnancy test | * | | | | | |



| Immunological evaluation (Saint-Antoine) | * | * | | | * | * |
|----------------------------------------------|----|----|---|---|---|---|
| Pharmacokinetic evaluation | | *6 | | | | |
| Pulmonary function test (FEV1) | * | | | | * | * |
| Chest x-ray | * | | | | | |
| Cutaneous biopsy (if relevant) | * | | | | | |
| ATO treatment (date, dose, reason of change) | | * | | | | |
| Response to treatment | | | | | * | |
| Associated treatment(s)8 | *7 | * | * | * | * | * |
| Adverse event(s) | | * | * | * | * | * |

<sup>&</sup>lt;sup>1</sup> During ATO treatment, must be performed daily before each ATO administration.

<sup>&</sup>lt;sup>2</sup> Must be performed weekly.

 $<sup>^{3}</sup>$  CBC included leucocytes, neutrophils, lymphocytes, monocytes, and eosinophils counts, hemoglobin and platelets.

<sup>&</sup>lt;sup>4</sup> Biochemistry included measurement of glycaemia<sup>9</sup>, creatinine<sup>1</sup>, uric acid, calcium<sup>1</sup>, potassium<sup>1</sup>, magnesium<sup>1</sup>, total protein, albumin, total bilirubin, alkaline phosphatases, SGOT<sup>9</sup>, SGPT<sup>9</sup>, and

<sup>&</sup>lt;sup>5</sup> Prothrombin time [PT], activated partial thromboplastin time [APTT].

<sup>&</sup>lt;sup>6</sup> Pharmacokinetic evaluation: the samples must be performed before each administration at D2, D3, D4, D5, D8, D12, D17 and D24 of cycle 1 and cycle 2 (if applicable).

 $<sup>^7</sup>$  History of GvHD prophylaxis : documentation of any associated treatments and topical therapy since graft for acute GvHD or progressive form of cGvHD treated by corticotherapy < 1 mg/kg/day, whenever possible given collected clinical history

<sup>&</sup>lt;sup>8</sup> Documentation of any associated treatments and topical therapy for chronic GvHD (including glucocorticoid creams, topical tacrolimus, oral beclomethasone or budesonide, topical azathioprine and ophthalmic glucocorticoids...)

<sup>&</sup>lt;sup>9</sup> Must be performed twice a week.

<sup>10</sup> Documentation on the diagnosis of hemopathy requiring transplant and DLI modality.




### 9.5 DATA QUALITY ASSURANCE

#### 9.5.1 GOOD CLINICAL PRACTICE

The study will be performed according to the Guidelines for Good Clinical Practice (ICH Harmonized Tripartite Guideline for Good Clinical Practice, (17.01.1997)).

The investigator will be thoroughly familiar with the appropriate use of the study drug as described in the protocol and SPC. Essential clinical documents will be maintained to demonstrate the validity of the study and the integrity of the data collected. A trial master file should be established at the beginning of the study, maintained for the duration of the study and retained according to the appropriate regulations.

#### 9.5.2 AUDITING

To guarantee a high quality of treatment for the patients within the present study, the sponsor will insure that the participating centres fulfill the following criteria:

- Fulfilling of legal requirements \_ experience of the principle investigator of the entire study and the respective centre with respect to study conduct
- International Conference on Harmonization (ICH)/GCP knowledge and certifications

#### 9.5.3 MONITORING

Regular monitoring is an essential part of the study conduct. It will be performed by the Sponsor of the study. After the initiation visit, the frequency of monitoring visits will depend on the course of the study, and recruitment. It is the monitor's responsibility to make the local investigators and all the staff who is involved into the study or the care of the patients familiar with the protocol.




During the course of the study, the monitor will control the progress of the study, the commitment to the protocol, the documentation and careful usage of the study medication, and the maintenance of GCP guidelines and legal obligations. Problems as well as changes in reported data will be worked out in collaboration with the local investigator, who is obliged to cooperate with the monitor and to allow access to the patients' charts. Source data verification is performed by the monitor. This protocol is classified as a "D" risk level estimated for the patients (Phase 11= very high risk predictable).

Inclusion criteria will be verified in 100% of patients. The monitor will have to respect that the data she/he comes into contact with are highly confidential. A monitoring report will be provided for each visit.

#### 9.5.4 DATA MANAGEMENT

The coding and data control for the exploitation of results of the study will be conducted by the Contract research Organization (CRO) in charge of the study, FOVEA (RueilMalmaison, France), according to its standard operating procedures, ICH guidelines, and under the supervision of the Sponsor.

#### 9.5.4.1 Data entry

All study data will be recorded and stored in a computerized database within the CRO, under the supervision of the Data Manager and under appropriate procedures. The data are available within the system to the Sponsor as soon as they are entered in the e-CRF.

#### 9.5.4.2 Consistency checks

Procedures for control of electronic data (Data Computer Management) will be defined to ensure the validity of information gathered as part of this study. They will cover all of the data and will aim to highlight abnormalities as missing data or inconsistent data.




These controls will be fully described in a manual of Data Management and will be implemented in the e-CRF. The computerized handling of the data by the Sponsor may generate additional requests (discrepancy resolution forms) to which the Investigator is obliged to respond by confirming or modifying the data questioned. The requests with their responses will be managed through the e-CRF.

### 9.5.4.3 Data coding

The AES will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), while previous treatments will be coded using the World Health Organization (WHO) dictionary according to anatomic-therapeutic-chemical classification (ATC).




# 12.4 STATISTICAL ANALYSIS METHODES PLANNED IN THE PROTOCOL AND DETERMINATION OF SAMPLE SIZE

#### 12.4.3 Statistical and Analytical Plans

#### 12.4.3.1 General approaches

All continuous data will be summarized using the following statistics: n (non-missing sample size), mean, standard deviation, median, minimum (min) and maximum (max). All categorical/qualitative data will be presented using the frequency and the percentage of patients who are in the particular category. In general, all data will be listed, sorted by site, subject, and by visit number within subject. All summary tables will be annotated with the total population size relevant to that table/treatment, including any missing observation.

The mean and the standard deviation will be reported to one decimal place greater than the original data. Median, minimum and maximum will use the same number of decimal places as the original data. P-values ≥0.001 will be reported to 3 decimal places; p-values less than 0.001 will be reported as "<0.001".

Type 1 error rate will be set at 0.05.

All statistical analyses will be conducted using SAS version 9.4.

#### 12.4.3.2 Handling of Dropouts or Missing Data

Every effort will be made to keep the number of missing values for all parameters to a minimum. The number of missing values will be reported together with summary statistics for each variable.

Missing data on overall survival is assumed to be null as patient care after transplantation is very close. Any patient prematurely withdrawn or ending the study without the event of interest (progression, death) will be censored at his/her last information date.

Concerning the main endpoint (response at M6), the missing assessments will be fully discussed during the data review. The most plausible outcome (the clinically more relevant) will be used for the main analysis. Other methods of imputation (for example, worst




outcome: missing data=failure) could be used for sensitivity purpose, according to the final number of missing assessments.

## 12.4.3.3 Interim Analyses

No interim analysis is planned.

### 12.4.3.4 Statistical analyses

A descriptive analysis will be conducted on the following parameters:

- Patients and transplant characteristics
- Primary and secondary endpoints

The toxicities rate will be calculated and will be given with their 95% confidence intervals.

The probabilities of survival will be estimated by the Kaplan-Meier method and by calculating the cumulative incidences for relapse/progression, and non-relapse mortality incidence.

#### 12.4.3.5 Determination of sample size

The aim of this study is to assess whether ATO allows improving response rate at 6 months after the diagnosis of chronic GVHD from 60% to 85%.

For the sample size calculation in this trial, an A'Hern one stage design has been used (ref 1).

- Let P0 be the smallest response rate, if true, implies that the role of ATO is too low and therefore the present schedule does not warrant further investigation. In the present trial, P0 has been taken as 60%.
- Let P1 be the highest response rate which, if true, implies that the feasibility is sufficiently high and therefore the current schedule warrants further investigation in clinical trials. In the present trial, P1 has been taken as 85%;
- Let  $\alpha$  be the accepted probability of recommending for further investigation a regimen with a true discontinuation rate at least equal to P0. In the present trial,  $\alpha$  has been taken as 0.05.
- Let  $\beta$  be the accepted probability of rejecting for further investigation a regimen with a true discontinuation rate less than P1. In the present trial,  $\beta$  has been taken as 0.20.




The required number of eligible patients is 21. To compensate for a dropout of 10%, 24 patients are planned to be included.

### 12.5 CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSIS

Any changes to the analyses described in the protocol or in approved versions of this plan will be fully documented in a specific part of the clinical study report of the study.




## 10.PATIENTS

## 10.1 DISPOSITION OF PATIENTS

All patients screened and receiving at least one infusion of ATO will be accounted for.

## **Derivation**

| Derived variables | Definition |
|-------------------|-------------------------------------------------------|
| Study completed | Yes, if the patient is present in the study at M12 |
| | No, if the patient is not present in the study at M12 |

The following table will be then presented:

| | Analysis set<br>(N=XX) |
|---|---|
| Study completed | n/N (XX.XX%) |
| Withdrawal of informed consent | n/N (XX.XX%) |
| Lost to follow-up | n/N (XX.XX%) |
| Occurrence of AE/SAE requiring premature discontinuation | n/N (XX.XX%) |
| Inclusion criteria not met requiring premature discontinuation | n/N (XX.XX%) |
| Other reason | n/N (XX.XX%) |




## 10.2 PROTOCOL DEVIATIONS

Protocol deviations will be summarized as follows:

## Analysis set (N=XX)

| | Number of patients | Number of deviations |
|-----------------|--------------------|----------------------|
| No deviation | n/N (XX.XX%) | n |
| Major deviation | n/N (XX.XX%) | n |




#### 11.EFFICACY EVALUATION

#### 11.1 ANALYSES POPULATIONS

Every patient included in the study and who has received at least one infusion of ATO will be taken into account at time of data analysis.

The number of patients included who did not receive any infusion of ATO will be reported as well as the reason for not receiving ATO.

The following analyses populations will be considered:

- The safety population consists of all patients included in the study for whom there is any evidence that they used at least one ATO injection.
- The Full Analysis Set (FAS) population consists of included subjects who completed their first cycle of ATO and for whom the response at Week 6 after diagnosis of chronic GvHD has been evaluated.
- The Per Protocol (PP) population will exclude FAS patients with any major protocol deviations that may impact the efficacy analysis. The exclusion of patients from the PP population will be determined during the final data review meeting. Reason(s) for exclusion will be documented for each patient.

The following table will be presented:

| Analysis<br>(N=XX | |
|------------------------------|--------------|
| Safety Population | n/N (XX.XX%) |
| Full Set Analysis Population | n/N (XX.XX%) |
| Per Protocol Population | n/N (XX.XX%) |




## 11.2 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

## 11.2.1 Demographic characteristics

## **Derivation**

| Derived variable | Definition |
|-----------------------------|-----------------------------------|
| Age at inclusion (in years) | Year of inclusion – Year of birth |

The following table will be presented:

| Variable | Statistics / Modality | Safety Population<br>(N = XX) |
|---|---|---|
| Gender | Male<br>Female<br>Missing | n/N (XX.X%)<br>n/N (XX.X%)<br>n |
| Age at inclusion (in years) | N (N Missing)<br>Mean ± SD<br>Median [Min ; Max] | XX (XX)<br>XX.X ± XX.X<br>XX [XX ; XX] |
| Contraception | Yes<br>No<br>Missing | n/N (XX.X%)<br>n/N (XX.X%)<br>n |
| Weight (kg) | N (N Missing)<br>Mean ± SD<br>Median [Min ; Max] | XX (XX)<br>XX.X ± XX.X<br>XX [XX ; XX] |
| Height (cm) | N (N Missing)<br>Mean ± SD<br>Median [Min ; Max] | XX (XX)<br>XX.X ± XX.X<br>XX [XX ; XX] |
| Cardiac frequency (beats/min) | N (N Missing)<br>Mean ± SD<br>Median [Min ; Max] | XX (XX)<br>XX.X ± XX.X<br>XX [XX ; XX] |
| Systolic arterial pressure (mmHg) | N (N Missing)<br>Mean ± SD<br>Median [Min ; Max] | XX (XX)<br>XX.X ± XX.X<br>XX [XX ; XX] |
| Diastolic arterial pressure (mmHg) | N (N Missing)<br>Mean ± SD<br>Median [Min ; Max] | XX (XX)<br>XX.X ± XX.X<br>XX [XX ; XX] |




| Temperature (°C) | N (N Missing) | XX (XX) |
|--------------------|--------------------|-----------------|
| | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| O2 activistics (%) | N (N Missing) | XX (XX) |
| O2 saturation (%) | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |

## 11.2.2 Baseline characteristics

## **Derivation**

| Derived variable | Definition |
|---|---|
| Time from transplant to chronic GVHD (in | Assessment date - Date of the first |
| days) | allogeneic stem cell transplantation +1 |
| Daily steroid dose (Prednisone): mg/kg/d | Considering the treatment line when the |
| | baseline occurs, the daily dose is calculated as: |
| | Dose*frequency/weight |
| | The frequency can be: once a day, twice a day, 1 day on 2 etc. |
| Daily cyclosporine dose | Considering the treatment line when the baseline occurs, the daily dose is |
| | calculated as: |
| | Dose*frequency |
| | The frequency can be: once a day, twice a day, 1 day on 2 etc. |




## The following table will be presented:

| Variable | Statistics / Modality | Safety Population<br>(N = XX) |
|---|---|---|
| | No | n/N (XX.X%) |
| Significant current disease | Yes | n/N (XX.X%) |
| | Missing | n |
| | Modality 1 | n/N (XX.X%) |
| Donor / Recipient features | Modality 2 | n/N (XX.X%) |
| | Modality n | n/N (XX.X%) |
| | Missing | n |
| Conditioning regimen | | |
| | Modality 1 | n/N (XX.X%) |
| Conditioning regimen | Modality 2 | n/N (XX.X%) |
| | Modality n | n/N (XX.X%) |
| | Missing | n |
| Previous infusion of DLI | | |
| DLI | No | n/N (XX.X%) |
| DEI | Yes | n/N (XX.X%) |
| | Missing | n |
| Time from transplant to G | | |
| Time from transplant to | N (N Missing) | XX (XX) |
| chronic GVHD (in days) | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Concomitant disease | | |
| Current disease? | No | n/N (XX.X%) |
| Current disease: | Yes | n/N (XX.X%) |
| | Missing | n |
| Haematology | | |
| | N (N Missing) | XX (XX) |
| Leucocytes | Mean ± SD | $X.XX \pm X.XX$ |
| · | Median [Min ; Max] | X.X [X.X ; X.X] |
| | N (N Missing) | XX (XX) |
| Neutrophils | Mean ± SD | $X.XX \pm X.XX$ |
| | Median [Min ; Max] | X.X [X.X ; X.X] |
| | N (N Missing) | XX (XX) |
| Lymphocytes | Mean ± SD | $X.XX \pm X.XX$ |
| | Median [Min ; Max] | X.X [X.X ; X.X] |



| | N (N Missing) | XX (XX) |
|---|---|---|
| Monocytes | Mean ± SD | $X.XX \pm X.XX$ |
| | Median [Min ; Max] | X.X [X.X ; X.X] |
| | N (N Missing) | XX (XX) |
| Eosinophils | Mean ± SD | $X.XX \pm X.XX$ |
| · | Median [Min ; Max] | X.X [X.X ; X.X] |
| | N (N Missing) | XX (XX) |
| Hemoglobin | Mean ± SD | $XX.XX \pm XX.XX$ |
| | Median [Min ; Max] | XX.X [XX.X ; XX.X] |
| | N (N Missing) | XX (XX) |
| Platelets | Mean ± SD | $XXX.X \pm XXX.X$ |
| | Median [Min ; Max] | XXX [XXX ; XXX] |
| aPTT | N (N Missing) | XX (XX) |
| агіі | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Serum chemistries | | |
| Creatinine | N (N Missing) | XX (XX) |
| Ordan mio | Mean ± SD | $XX.XX \pm XX.XX$ |
| | Median [Min ; Max] | XX.X [XX.X ; XX.X] |
| Uric acid | N (N Missing) | XX (XX) |
| | Mean ± SD | XXX.X ± XXX.X |
| | Median [Min ; Max] | XXX [XXX ; XXX] |
| Total bilirubin | N (N Missing)<br>Mean ± SD | XX (XX) |
| | | XX.XX ± XX.XX |
| | Median [Min ; Max] | XX.X [XX.X ; XX.X] |
| Alkaline phosphatases | N (N Missing)<br>Mean ± SD | XX (XX)<br>XXX.X ± XXX.X |
| | Median [Min ; Max] | XXX [XXX ; XXX] |
| | N (N Missing) | XX (XX) |
| LDH | Mean ± SD | $XXX.X \pm XXX.X$ |
| | Median [Min ; Max] | XXX [XXX ; XXX] |
| | N (N Missing) | XX (XX) |
| Total protein | Mean ± SD | XX.X ± XX.X |
| | Median [Min ; Max] | XX [XX ; XX] |
| | N (N Missing) | XX (XX) |
| Albumin | Mean ± SD | $XX.XX \pm XX.XX$ |
| | Median [Min ; Max] | XX.X [XX.X; XX.X] |
| SCOT | N (N Missing) | XX (XX) |
| SGOT | Mean ± SD | XXX.X ± XXX.X |
| | Median [Min ; Max] | XXX [XXX ; XXX] |



| SCDT | N (N Missing) | XX (XX) |
|--------------------------|----------------------------|--------------------|
| SGPT | Mean ± SD | $XXX.X \pm XXX.X$ |
| | Median [Min ; Max] | XXX [XXX ; XXX] |
| Calaium | N (N Missing) | XX (XX) |
| Calcium | Mean ± SD | $X.XXX \pm X.XXX$ |
| | Median [Min ; Max] | X.XX [X.XX ; X.XX] |
| Oh | N (N Missing) | XX (XX) |
| Glycaemia | Mean ± SD | X.XX ± X.XX |
| | Median [Min ; Max] | X.X [X.X ; X.X] |
| Infectious disease surv | | • |
| | Negative | n/N (XX.X%) |
| CMV | Positive | n/N (XX.X%) |
| | Missing | 'n |
| ED. / | Negative | n/N (XX.X%) |
| EBV | Positive | n/N (XX.X%) |
| | Missing | n , |
| | Negative | n/N (XX.X%) |
| Hepatitis B | Positive | n/N (XX.X%) |
| | Missing | n , |
| lmmunology | | |
| | N (N Missing) | XX (XX) |
| Gammaglobulin level | Mean ± SD | XX.XX ± XX.XX |
| | Median [Min ; Max] | XX.X [XX.X ; XX.X] |
| | Negative | n/N (XX.X%) |
| Antinuclear antibody | Positive | n/N (XX.X%) |
| | Missing | n |
| | Negative | n/N (XX.X%) |
| ANCA | Positive | n/N (XX.X%) |
| | Missing | n , |
| Cardiac assessment | 5 | |
| | Not realized | n/N (XX.X%) |
| EKG – Performed? | Realized | n/N (XX.X%) |
| | Missing | 'n |
| | Abnormal | n/N (XX.X%) |
| EKG – Result | Normal | n/N (XX.X%) |
| | Missing | n |
| | N (N Missing) | XX (XX) |
| QTc | Mean ± SD | XXX.X ± XXX.X |
| | Median [Min ; Max] | XXX [XXX ; XXX] |
| Serum levels of electrol | | 700([700(,700(] |
| | N (N Missing) | XX (XX) |
| Potassium | Mean ± SD | X.XX ± X.XX |
| | Median [Min ; Max] | X.X [X.X ; X.X] |
| Magnesium | N (N Missing) | XX (XX) |
| Magnosiani | 14 (14 1411331119 <i>)</i> | /V( /V() |



| | Mean ± SD | X.XXX ± X.XXX |
|---------------------------|--------------------|--------------------|
| | Median [Min ; Max] | X.XX [X.XX ; X.XX] |
| Results of other tests | - | - |
| | 0 | n/N (XX.X%) |
| | 1 | n/N (XX.X%) |
| Performance status | 2 | n/N (XX.X%) |
| | 3 | n/N (XX.X%) |
| | 4 | n/N (XX.X%) |
| | Missing | n |
| Karnafaky indov | N (N Missing) | XX (XX) |
| Karnofsky index | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Choot V ray | Not realized | n/N (XX.X%) |
| Chest X ray | Realized | n/N (XX.X%) |
| | Missing | n |
| If realized, chest X ray | Abnormal | n/N (XX.X%) |
| result | Normal | n/N (XX.X%) |
| | Missing | n |
| Cutanagua bianay | Not realized | n/N (XX.X%) |
| Cutaneous biopsy | Realized | n/N (XX.X%) |
| | Missing | n |
| If realized, cutaneous | Abnormal | n/N (XX.X%) |
| biopsy result | Normal | n/N (XX.X%) |
| | Missing | n |
| % FEV1 | N (N Missing) | XX (XX) |
| /0 F E V I | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Concomitant treatment | | |
| Any concomitant | No | n/N (XX.X%) |
| treatments administrated? | Yes | n/N (XX.X%) |
| | Missing | n |
| Daily steroid dose | N (N Missing) | XX (XX) |
| (Prednisone) | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| mg/kg/d | | |
| Daily cyclosporine dose | N (N Missing) | XX (XX) |
| Daily Cyclospolitic dose | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |




#### Signs and symptoms of cGvHD at baseline 11.2.3

## **Derivation**

| Derived variable | Definition |
|---|---|
| Liver score | The liver score is defined as a combination of Total bilirubin, ALT (SGPT) and AP (ALK) as follows: |
| | Score 0: Normal total bilirubin and ALT < 3 ULN and AP < 3 ULN |
| | Score 1: Normal total bilirubin with ALT ≥ 3 to 5 ULN or AP ≥ 3 to 5 ULN |
| | Score 2: Elevated total bilirubin (> 1 ULN) but ≤ 3 mg/dL or ALT ≥ 5 ULN or AP ≥ 5 ULN |
| | Score 3: Elevated total bilirubin > 3 mg/dL |
| | Missing if at least one missing serum chemistry |
| Involved sites number | Number of sites or organs with a score ≥ 1 at baseline (V1) |

The following table will be presented:

| Variable | Statistics / Modality | Safety Population<br>(N = XX) |
|---|---|---|
| NIH scoring of cGVHD | | |
| | Score 0: Asymptomatic and fully active (ECOG 0, KPS or LPS 100%) | n/N (XX.X%) |
| Scoring of chronic GVHD (NIH criteria) | Score 1: Symptomatic, fully ambulatory, restricted only in physically strenuous activity (ECOG 1, KPS or LPS 80-90 %) | n/N (XX.X%) |
| | Score 2: Symptomatic ambulatory, capable of selfcare, | n/N (XX.X%) |



| | > 50 % of walking hours out of bed<br>(ECOG 2, KPS or<br>LPS 60-70 %) | |
|---|---|---|
| | Score 3: Symptomatic, limited self-<br>care > 50 % of<br>waking hours in bed (ECOG 3-4,<br>KPS or LPS < 60 %) | n/N (XX.X%) |
| | Missing | n |
| Skin – Abnormalities<br>present but explained | No | n/N (XX.X%) |
| entirely by non-GvHD<br>documented cause | Yes | n/N (XX.X%) |
| | Missing | n |
| | Score 0: No BSA involved | n/N (XX.X%) |
| | Score 1: 1-18% BSA | n/N (XX.X%) |
| Skin score | Score 2: 19-50% BSA | n/N (XX.X%) |
| | Score 3: > 50% BSA | n/N (XX.X%) |
| | Missing | n |
| Mouth – Abnormalities<br>present but explained | No | n/N (XX.X%) |
| entirely by non-GvHD<br>documented cause | Yes | n/N (XX.X%) |
| | Missing | n |
| | Score 0: No symptoms | n/N (XX.X%) |
| | Score 1: Mild symptoms with disease signs but not limiting oral intake significantly | n/N (XX.X%) |
| Mouth score | Score 2: Moderate symptoms with disease signs with partial limitation or oral intake | n/N (XX.X%) |
| | Score 3: Severe symptoms with disease signs on examination with | n/N (XX.X%) |
| | major limitation or oral intake | |



| Lung – Abnormalities | No | n/N (XX.X%) |
|---|---|---|
| present but explained<br>entirely by non-GvHD<br>documented cause | Yes | n/N (XX.X%) |
| documented cause | Missing | n |
| | Score 0: No symptoms | n<br>n/N (XX.X%) |
| Lung score + FEV1 | Score 1: Mild symptoms (shortness of breath after climbing one flight of steps) Score 2: Moderate symptoms (shortness of breath after walking on flat ground) | n/N (XX.X%)<br>n/N (XX.X%) |
| | Score 3: Severe symptoms (shortness of breath at rest: requiring 0) | n/N (XX.X%) |
| | NAI | n |
| Fyee Abnormalities | Missing | ~/N /VV V0/ \ |
| Eyes – Abnormalities present but explained | No | n/N (XX.X%) |
| entirely by non-GvHD<br>documented cause | Yes | n/N (XX.X%) |
| documented dauge | Missing | n |
| | Score 0: No symptoms | n/N (XX.X%) |
| | Score 1: Mild dry eye symptoms not affecting ADL | n/N (XX.X%) |
| Eyes score | Score 2: Moderate dry eye symptoms partially affecting ADL without new vision impairment due to KCS | n/N (XX.X%) |
| | Score 3: Severe eye symptoms significantly affecting ADL or unable to work because of ocular | n/N (XX.X%) |
| | symptoms of loss or vision due to KCS | n |
| | Missing | |
| | No | n/N (XX.X%) |
| Gastro-intestinal –<br>Abnormalities present but | Yes | n/N (XX.X%) |



| explained entirely by non-<br>GvHD documented cause | Missing | n |
|---|---|---|
| | Score 0: No symptoms | n/N (XX.X%) |
| | Score 1: Symptoms without significant weight loss (< 5 %) | n/N (XX.X%) |
| Gastro-intestinal score | Score 2: Symptoms associated with mild to moderate weight loss (5-15%) OR moderate diarrhea without significant interference with daily living | n/N (XX.X%) |
| | Score 3: Symptoms associated with significant weight loss > 15 %, requires nutritional supplement for most calorie needs OR esophageal dilation OR severe diarrhea with significant interference with daily living | n/N (XX.X%) |
| | Missing | n |
| Liver – Abnormalities present but explained | No | n/N (XX.X%) |
| entirely by non-GvHD<br>documented cause | Yes | n/N (XX.X%) |
| | Missing | n |
| | Score 0: Normal total bilirubin and ALT or AP < 3 ULN | n/N (XX.X%) |
| | Score 1: Normal total bilirubin with ALT ≥ 3 to 5 ULN and AP ≥ 3 to 5 ULN | n/N (XX.X%) |
| Liver score | Score 2: Elevated total bilirubin (> 1 ULN) but ≤ 3 mg/dL or ALT ≥ 5 ULN or AP ≥ 5 ULN | n/N (XX.X%) |
| | Score 3: Elevated total bilirubin > 3 mg/dL | n/N (XX.X%) |
| | Missing | n |
| Joint and fascia –<br>Abnormalities present but | No | n/N (XX.X%) |



| avalained entirely by nen | Vac | n/NI /VV V0/ \ |
|---|---|---|
| explained entirely by non-<br>GvHD documented cause | Yes | n/N (XX.X%) |
| GVID documented cause | Missing | n |
| | Score 0: No symptoms | n/N (XX.X%) |
| | Ocore of two symptoms | 11/14 (704.7470) |
| | Score 1: Mild tightness of arms or legs, normal or mild decreased range of motion (ROM) AND not affecting ADL | n/N (XX.X%) |
| | | n/N (XX.X%) |
| Joints and fascia score | Score 2: Tightness of rams and legs OR joints contractures, erythema thought due to fasciitis, moderate decrease ROM AND mild to moderate limitation of ADL | n/N (XX.X%) |
| | Score 3: Contractures WITH significant decrease of ROM AND significant limitation of ADL (unable to tie shoes, button shirts, dress self, etc) | |
| | Missing | n |
| Involved sites number | | |
| Involved sites number | N (N Missing) | XX (XX) |
| involved sites number | Mean ± SD | $X.X \pm X.X$ |
| | Median [Min ; Max] | X [X ; X] |
| Current patient weight | | |
| Current patient weight (in | N (N Missing) | XX (XX) |
| kg) | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Performance score | | |
| | KPS | n/N (XX.X%) |
| Performance status | ECOG | n/N (XX.X%) |
| | LPS | n/N (XX.X%) |
| | Missing | n |
| | ECOG 1 | n/N (XX.X%) |
| If ECOG | ECOG 2 | n/N (XX.X%) |
| | ECOG 3 | n/N (XX.X%) |
| | Missing | n |
| Chronic GVHD activity as | | ••• |
| Overall GvHD severity | No GVHD | n/N (XX.X%) |
| 2.3.a. 21.12 001011tg | · | \ |
| | Mild | n/N (XX.X%) |



| | Moderate | n/N (XX.X%) |
|-------------------------|---------------------|-----------------|
| | Severe | n/N (XX.X%) |
| | Missing | n |
| Assessment of cGVHD | N (N Missing) | XX (XX) |
| severity (from 0 to 10) | Mean ± SD | $XX.X \pm XX.X$ |
| • . | Median [Min ; Max] | XX [XX ; XX] |
| Chronic GVHD activity a | ssessment - Patient | |
| Assessment of cGVHD | N (N Missing) | XX (XX) |
| severity (from 0 to 10) | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |




## 11.3 ATO AND ASSOCIATED TREATMENTS

## 11.3.1 Arsenic trioxide therapy

## **Derivation**

| Derived variables | Definition |
|---|---|
| Time from diagnosis of cGvHD to first infusion of ATO (in days) | Date of Cycle 1 onset – GvHD assessment date + 1 |
| The same derivation will be applied for each ATO infusion | Missing if one of the two dates is missing |
| Time from starting Prednisone to first infusion of ATO (in days) | Date of Cycle 1 onset – Date of<br>Prednisone onset +1 |
| | Missing if one of the two dates is missing |
| Number of cycles | 1, if a date of cycle 1 onset is known |
| | 2, if a date of cycle 2 onset is known |
| | Missing otherwise |
| Total dose during Wi | For the considered period (Wi), sum of each dose took |
| Calculated at Wi={W1, W2, W3, W4} of each cycle | Example: C1_D1+C1_D2+C1_D3+C1_D5 for the first week |
| Daily dose during Wi | For the considered week, the daily dose will be calculated as follows: |
| Calculated at Wi={W1, W2, W3, W4} of each cycle | Total dose / Number of days with intake treatment during Wi |
| Time from the first infusion of ATO to the first day of the second cycle (in days) | Date of Cycle 2 onset – Date of Cycle 1 +1 Missing if one of the two dates is missing |
| Temporary discontinuation of ATO | Yes, if at least one missing infusion during the cycle 1 or cycle 2 if initiated |




| No, if the patient has received all the planned doses |
|-------------------------------------------------------|

## The following table will be presented:

| Variable | Statistics / Modality | Safety Population<br>(N = XX) |
|---|---|---|
| Time from diagnosis of | N (N Missing) | XX (XX) |
| cGvHD to first infusion of | Mean ± SD | $XX.X \pm XX.X$ |
| ATO (in days) | Median [Min ; Max] | XX [XX ; XX] |
| Time from diagnosis of | N (N Missing) | XX (XX) |
| cGvHD to second infusion | Mean ± SD | $XX.X \pm XX.X$ |
| of ATO (in days) | Median [Min ; Max] | XX [XX ; XX] |
| Time from diagnosis of | N (N Missing) | XX (XX) |
| cGvHD to last infusion of | Mean ± SD | $XX.X \pm XX.X$ |
| ATO (in days) | Median [Min ; Max] | XX [XX; XX] |
| Time from starting | N (N Missing) | XX (XX) |
| Prednisone to first infusion | Mean ± SD | $XX.X \pm XX.X$ |
| of ATO (in days) | Median [Min ; Max] | XX [XX; XX] |
| Number of quality | 1 | n/N (XX.X%) |
| Number of cycles | 2 | n/N (XX.X%) |
| | Missing | n |
| First cycle | | 201.000 |
| Number of infusions | N (N Missing) | XX (XX) |
| | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Number of weeks | N (N Missing) | XX (XX) |
| | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Week 1 | | 207.000 |
| Daily dose during W1 | N (N Missing) | XX (XX) |
| =, | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Number of days during W1 | N (N Missing) | XX (XX) |
| | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Total dose during W1 | N (N Missing) | XX (XX) |
| | Mean ± SD | XX.X ± XX.X |



| | Median [Min ; Max] | XX [XX ; XX] |
|------------------------------|--------------------|-----------------|
| Week 2 | , | , , |
| Doily does during M2 | N (N Missing) | XX (XX) |
| Daily dose during W2 | Mean ± SD | XX.X ± XX.X |
| | Median [Min ; Max] | XX [XX ; XX] |
| Number of days during W2 | N (N Missing) | XX (XX) |
| Number of days during W2 | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Total daga during W2 | N (N Missing) | XX (XX) |
| Total dose during W2 | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Week 3 | | |
| Daily dose during W3 | N (N Missing) | XX (XX) |
| Daily dose during W3 | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Number of days during W3 | N (N Missing) | XX (XX) |
| Number of days during wo | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Total dose during W3 | N (N Missing) | XX (XX) |
| Total dose during W3 | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Week 4 | | |
| Daily dose during W4 | N (N Missing) | XX (XX) |
| Daily dose during W4 | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Number of days during W4 | N (N Missing) | XX (XX) |
| Number of days during VV+ | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Total dose during W4 | N (N Missing) | XX (XX) |
| Total dose during W+ | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Temporary discontinuation | No | n/N (XX.X%) |
| of ATO* | Yes | n/N (XX.X%) |
| | Missing | n |
| Second cycle | | |
| Patients who entered into | No | n/N (XX.X%) |
| the 2 <sup>nd</sup> cycle | Yes | n/N (XX.X%) |
| | Missing | n |
| Time from the first infusion | N (N Missing) | XX (XX) |
| of ATO to the first day of | Mean ± SD | $XX.X \pm XX.X$ |
| the second cycle (in days) | Median [Min ; Max] | XX [XX ; XX] |
| Number of infusions | N (N Missing) | XX (XX) |
| 140/1100/ OF HITUSIONS | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |



| Week 1 | | |
|-------------------------------|--------------------|-----------------|
| Daile da a demis e MA | N (N Missing) | XX (XX) |
| Daily dose during W1 | Mean ± SD | XX.X ± XX.X |
| | Median [Min ; Max] | XX [XX ; XX] |
| Number of days during 1974 | N (N Missing) | XX (XX) |
| Number of days during W1 | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Total dage during W/1 | N (N Missing) | XX (XX) |
| Total dose during W1 | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Week 2 | | |
| Daily dose during W2 | N (N Missing) | XX (XX) |
| Daily dose during W2 | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Number of days during W2 | N (N Missing) | XX (XX) |
| Number of days during W2 | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Total dose during W2 | N (N Missing) | XX (XX) |
| rotal dose during wz | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Week 3 | | |
| Daily dose during W3 | N (N Missing) | XX (XX) |
| Daily dose during wo | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Number of days during W3 | N (N Missing) | XX (XX) |
| Number of days during W5 | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Total dose during W3 | N (N Missing) | XX (XX) |
| Total dose during Wo | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Week 4 | | |
| Daily dose during W4 | N (N Missing) | XX (XX) |
| Bany door daring W | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Number of days during W4 | N (N Missing) | XX (XX) |
| realiser of days dailing vv i | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Total dose during W4 | N (N Missing) | XX (XX) |
| rotal doos daming Tr | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Temporary discontinuation | No | n/N (XX.XX%) |
| of ATO | Yes | n/N (XX.XX%) |
| | Missing | n |




In case of temporary discontinuation of ATO, a listing will be provided.




#### 11.3.2 Associated treatment

## • Prednisone and Ciclosporin A

## **Derivation**

| Derived variables | Definition |
|---|---|
| Time from diagnosis of cGvHD to Prednisone onset (in days) | Date of Prednisone onset – GvHD assessment date +1 Missing if one of the two dates is missing |
| Time from diagnosis of cGvHD to Ciclosporin onset (in days) | Date of Ciclosporin onset – GvHD assessment date +1 Missing if one of the two dates is missing |
| Treatment duration (in days) Calculated for Prednisone and Ciclosporin | Last treatment line end date – First treatment line start date +1 Missing if one of the two dates is missing |
| Daily dose for Prednisone and Ciclosporin Calculated for Prednisone (mg/kg/d) and Ciclosporin (mg/d) separately | First, for each treatment line, the total dose will be calculated as follows: dose*frequency*number of days The frequency can be: once a day, twice a day, 1 day on 2 etc. The average daily dose is then defined as follows: Sum of each dose treatment line / Treatment duration |
| Reason of change | As the treatment of a same patient can be changed several times, if a reason of change is met more than once, it will only be counted as one reason. Thus, the denominator will be the same as the analysis population (i.e. Safety Population) |




| - 1 | Secondary immunosuppressive treatment after first ATO infusion | No, if no treatment intake |
|---|---|---|
| | atel ilist ATO iliusion | Yes, if at least one treatment intake |

The following table will be presented:

| Variable | Statistics / Modality | Safety Population<br>(N = XX) |
|---|---|---|
| Prednisone | | , , |
| Time from diagnosis of | N (N Missing) | XX (XX) |
| cGvHD to first Prednisone | Mean ± SD | $XX.X \pm XX.X$ |
| dose (in days) | Median [Min ; Max] | XX [XX ; XX] |
| Treatment duration (in | N (N Missing) | XX (XX) |
| days) | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Daily dose (mg/kg/d) | N (N Missing) | XX (XX) |
| Daily dose (Hig/kg/d) | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Number of changes | N (N Missing) | XX (XX) |
| Number of changes | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| | Reason 1 | n/N (XX.X%) |
| Reason of change | Reason 2 | n/N (XX.X%) |
| | <br>Reason n | n/N (XX.X%) |
| Ciclosporin | | |
| Ciolognaria intaka | No | n/N (XX.X%) |
| Ciclosporin intake | Yes | n/N (XX.X%) |
| | Missing | n |
| Time from diagnosis of | N (N Missing) | XX (XX) |
| cGvHD to first Ciclosporin | Mean ± SD | $XX.X \pm XX.X$ |
| dose (in days) | Median [Min ; Max] | XX [XX ; XX] |
| Treatment duration (in | N (N Missing) | XX (XX) |
| days) | Mean ± SD | $XX.X \pm XX.X$ |
| - | Median [Min ; Max] | XX [XX ; XX] |
| Doily doos (mg/d) | N (N Missing) | XX (XX) |
| Daily dose (mg/d) | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| Number of changes | N (N Missing) | XX (XX) |
| Number of changes | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |




| Reason of change | Reason 1<br>Reason 2 | n/N (XX.X%)<br>n/N (XX.X%) |
|------------------|----------------------|----------------------------|
| | <br>Reason n | n/N (XX.X%) |

## • Concomitant treatments

Concomitant treatments will be presenting by descending sort of use.

The following table will be presented:

| | Safety Population<br>(N=XX) |
|---|---|
| Patients who received at least one concomitant treatment | n/N (XX.X%) |
| TRT 1 | n/N (XX.X%) |
| TRT 2 | n/N (XX.X%) |
| TRT n | <br>n/N (XX.X%) |

## • Secondary immunosuppressive treatment

| Variable | Statistics / Modality | Safety Population<br>(N = XX) |
|-------------------|-----------------------|-------------------------------|
| Secondary | No | n/N (XX.X%) |
| immunosuppressive | Yes | n/N (XX.X%) |
| treatment | Missing | n |




### 11.4 EFFICACY ANALYSIS

## 11.4.1 Primary Endpoint analysis

## 11.4.1.1 Response at 6 months – Main analysis

## • Complete or Partial response at 6 months (PI response)

The proportion of response at 6 months (CR or PR) will be estimated and presented with its 95% exact (Clopper-Pearson) confidence interval. The null hypothesis H0:  $P \le P0$  will be rejected in favor of the alternative hypothesis H1:  $P \ge P1$  if the lower bound of the 95% CI is lower than 60%.

#### **Derivation**

| Derived variables | Definition |
|---|---|
| Complete or partial response | Yes, if the PI judged the patient in complete or partial response at M6 |
| | No otherwise |

#### The following table will be presented:

| Variable | Modality | FAS Population (N = XX) |
|----------------|------------------------------|-------------------------|
| Response at M6 | Complete or partial response | n/N (XX.X%) [95% CI] |




#### • Complete and Partial response at 6 months (PI response)

Proportion of CR and PR at 6 months will also be estimated separately, and presented with their 95% exact (Clopper-Pearson) confidence intervals.

The following table will be presented:

| Variable | Modality | FAS Population<br>(N = XX) |
|---|---|---|
| Response at M6 | Complete response Partial response | n/N (XX.X%) [95% CI]<br>n/N (XX.X%) [95% CI] |

Responses and their 95% CI will be graphically represented using a forest plot.

Furthermore, previous analyses will be performed considering the following subgroups:

- By sex
- By center
- By number of cycles of ATO (1 or 2)
- By use of Ciclosporin or not
- By number of organs involved in cGvHD
- By GvHD severity at baseline

# 11.4.1.2 Response at 6 months – Sensitivity analyses

- a) The analysis presented in §11.4.1.1 will be performed on PP population
- b) The analysis presented in §11.4.1.1 will be performed on the response at 6 months computed by Soladis.
- c) The analysis presented in §11.4.1.1 will be performed on the response at 6 months based on the PI response, but excluding patients 06-07, 06-08 and 06-09.
- d) The analysis presented in §11.4.1.1 will be performed on the response at 6 months computed by Soladis, but excluding patients 06-07, 06-08 and 06-09.




## 11.4.2 Secondary Endpoint analyses

## 11.4.2.1 Response by organ

The proportion of response at 6 months (Complete, partial or progressive) will be estimated and presented for each organ. No response is evaluated for an organ when no abnormalities is present at V1, except progressive disease.

### **Derivation**

| Derived variables | Definition |
|----------------------------------|-------------------------------------------|
| Complete response for each organ | |
| Partial response for each organ | Cf Appendix 1 "Evaluation de la réponse – |
| Progressive disease | 19OCT2020" |
| Organ not involved at any moment | |

The following table will be presented:

| Organ | Response at M6 | FAS Population<br>(N = XX) |
|---|---|---|
| Organ 1 | Complete response Partial response | n/N (XX.X%)<br>n/N (XX.X%) |
| | Progressive disease Organ not involved at any moment | n/N (XX.X%)<br>n/N (XX.X%) |

This table will be completed for skin, mouth, lung, eyes, gastro-intestinal, liver and joint & fascia.




## 11.4.2.2 Survival analyses

## a) Failure free survival

A survival analysis will be conducted to describe the occurrence of failure between the first infusion of ATO and Vi, with Vi={M6;M12}.

### **Derivation**

| Derived variables | Definition |
|---|---|
| Failure at Vi | Defined as death, recurrent or progressive malignancy, or the initiation of a new |
| Calculated at Vi={M6;M12} | systemic treatment for chronic GvHD. |
| | Systemic treatment are: Methotrexate, Rapamune, TLI, Extracorporeal |
| | photopheresis, Rituximab, Jakavi, Glivec, |
| | Prograf, Imurel or other medications specified into the CRF (Vi RESP FAIL |
| | and or Vi_RESP_FAIL_S) |
| Time calculation from first ATO infusion to | If the event appears: the difference of date |
| failure at Vi | between the first ATO infusion and the first failure (expressed in months) is calculated. |
| Calculated at Vi={M6;M12} | The event will be not censured. |
| | (Date of first ATO infusion – Date of first failure)/30.5 |
| | If the event does not appear, the difference of date between the first ATO infusion and Vi (expressed in months) is |
| | infusion and Vi (expressed in months) is calculated. The event will be censured. |

The following table will be presented at M6:



| | | FAS Population |
|---|---|---|
| | | (N = XX) |
| First time of failure between first ATO infusion and M6 (in months) | n/M (%) of events | n/N (XX.XX%) |
| | n/M (%) of censored | n/N (XX.XX%) |

The Kaplan-Meier survival estimates will be plotted with the number of subjects at risk and 95% confidence limits.

These analyses will be also presented at M12.




#### b) Progression free survival

A survival analysis will be conducted to describe the occurrence of progression between the first infusion of ATO and Vi, with Vi={M6;M12}.

#### **Derivation**

| Derived variables | Definition |
|---|---|
| Progressive disease at Vi | Global progressive disease as define in Appendix 17.1 |
| Calculated at Vi={M6;M12} | |
| Time calculation from first ATO infusion to failure at Vi | If the event appears: the difference of date between the first ATO infusion and the first progression (expressed in months) is |
| Calculated at Vi={M6;M12} | calculated. The event will be not censured. |
| | (Date of first ATO infusion – Date of first progression)/30.5 |
| | If the event does not appear, the difference of date between the first ATO infusion and Vi (expressed in months) is calculated. The event will be censured. |

The following table will be presented at M6:

| | | FAS Population |
|---|---|---|
| | | (N = XX) |
| First time of progression between first ATO infusion and M6 (in months) | n/M (%) of events | n/N (XX.XX%) |
| | n/M (%) of censored | n/N (XX.XX%) |

The Kaplan-Meier survival estimates will be plotted with the number of subjects at risk and 95% confidence limits.

These analyses will be also presented at M12.




#### c) Overall survival

A survival analysis will be conducted to describe the occurrence of death between the first infusion of ATO and Vi, with Vi={M6;M12}.

## **Derivation**

| Derived variables | Definition |
|---|---|
| Death at Vi | Yes, if the death occurs between the first ATO infusion and Vi |
| Calculated at Vi={M6;M12} | |
| Time calculation from first ATO infusion to death at Vi | If the event appears: the difference of date between the first ATO infusion and the date of death (expressed in months) is |
| Calculated at Vi={M6;M12} | calculated. The event will be not censured. |
| | (Date of first ATO infusion – Date of death)/30.5 |
| | If the event does not appear, the difference of date between the first ATO infusion and Vi (expressed in months) is calculated. The event will be censured. |

The following table will be presented at M6:

| | | FAS Population |
|---|---|---|
| | | (N = XX) |
| Death between first ATO infusion and M6 (in months) | n/M (%) of events | n/N (XX.XX%) |
| | n/M (%) of censored | n/N (XX.XX%) |

The Kaplan-Meier survival estimates will be plotted with the number of subjects at risk and 95% confidence limits.

These analyses will be also presented at M12.




## 11.4.2.3 Treatment by Corticosteroids

## **Derivation**

| Derived variables | Definition |
|---|---|
| Selection of Prednisone treatment line at Vi | For each visit of interest, the Prednisone treatment line selected will be the one as: |
| Calculated for Vi = {W6, W14, M6, M9, M12} | Prednisone onset date ≤ Vi ≤ Prednisone end date |
| 1013, 10112j | If the visit matches with the Prednisone onset date, then the previous line is selected. |
| | If the visit matches with the Prednisone end date, then the current line is selected. |
| | If the visit cannot match with any treatment line then a missing value will be considered for this visit. |
| Daily dose for Prednisone at Vi | For each visit, the daily dose is calculated as: |
| Calculated for Vi = {W6, W14, M6, M9, M12} | dose*frequency/weight |
| 1V13, 1V112f | The frequency can be: once a day, twice a day, 1 day on 2 etc. |
| | Then the following categories will be created: |
| | ≤ 0.25 mg/kg/d |
| | 0.26 - 0.50 mg/kg/d |
| | 0.51 – 0.75 mg/kg/d |
| | 0.71 – 1 mg/kg/d |
| Change from baseline at Vi | Decreased, if dose category at Vi < dose category at baseline |
| Calculated for Vi = {W6, W14, M6, M9, M12} | Unchanged, if dose category at Vi = dose category at baseline |
| | Increased, if dose category at Vi > dose category at basleine |




| If the Prednisone treatment is not started at baseline then the date of first ATO infusion will be considered. |
|---|

The following table will be then presented:

| Visit | Variable | Statistics | FAS Population<br>(N=XX) |
|---|---|---|---|
| W6 | Daily dose for<br>Prednisone | ≤ 0.25 mg/kg/d<br>0.26 – 0.50 mg/kg/d<br>0.51 – 0.75 mg/kg/d<br>0.71 – 1 mg/kg/d<br>Missing | n/N (XX.XX%)<br>n/N (XX.XX%)<br>n/N (XX.XX%)<br>n/N (XX.XX%)<br>n |
| | Change from baseline | Decreased Unchanged Increased Missing | n/N (XX.XX%)<br>n/N (XX.XX%)<br>n/N (XX.XX%)<br>n |
| W14 | Daily dose for<br>Prednisone | ≤ 0.25 mg/kg/d<br>0.26 – 0.50 mg/kg/d<br>0.51 – 0.75 mg/kg/d<br>0.71 – 1 mg/kg/d<br>Missing | n/N (XX.XX%)<br>n/N (XX.XX%)<br>n/N (XX.XX%)<br>n/N (XX.XX%)<br>n |
| | Change from baseline | Decreased<br>Unchanged<br>Increased<br>Missing | n/N (XX.XX%)<br>n/N (XX.XX%)<br>n/N (XX.XX%)<br>n |
| M6 | Daily dose for<br>Prednisone | ≤ 0.25 mg/kg/d<br>0.26 – 0.50 mg/kg/d<br>0.51 – 0.75 mg/kg/d<br>0.71 – 1 mg/kg/d<br>Missing | n/N (XX.XX%)<br>n/N (XX.XX%)<br>n/N (XX.XX%)<br>n/N (XX.XX%)<br>n |
| Change from basel | Change from baseline | Decreased<br>Unchanged<br>Increased<br>Missing | n/N (XX.XX%)<br>n/N (XX.XX%)<br>n/N (XX.XX%)<br>n |
| M9 | Daily dose for<br>Prednisone | ≤ 0.25 mg/kg/d<br>0.26 – 0.50 mg/kg/d<br>0.51 – 0.75 mg/kg/d<br>0.71 – 1 mg/kg/d<br>Missing | n/N (XX.XX%)<br>n/N (XX.XX%)<br>n/N (XX.XX%)<br>n/N (XX.XX%)<br>n |
| | Change from baseline | Decreased<br>Unchanged<br>Increased | n/N (XX.XX%)<br>n/N (XX.XX%)<br>n/N (XX.XX%) |




| | | Missing | n |
|---|---|---|---|
| | Delhadasa fara | ≤ 0.25 mg/kg/d | n/N (XX.XX%) |
| | | 0.26 – 0.50 mg/kg/d | n/N (XX.XX%) |
| | Daily dose for | 0.51 - 0.75 mg/kg/d | n/N (XX.XX%) |
| Prednisone M12 Change from baseling | Prednisone | 0.71 – 1 mg/kg/d | n/N (XX.XX%) |
| | | Missing | 'n |
| | | Decreased | n/N (XX.XX%) |
| | Object of freeze becaling | Unchanged | n/N (XX.XX%) |
| | Change from baseline | Increased | n/N (XX.XX%) |
| | | Missing | 'n |

The daily dose for Prednisone over time and the change from baseline will be graphically represented by stacked bars.




## 11.4.2.4 Quality of life assessment

#### • FACT-BMT

## **Derivation**

| Derived variables | Definition |
|---|---|
| Physical well-being subscore at Vi | 7 * (Sum of the items GP1 to GP7) / Number of items answered |
| Calculated for Vi = {Baseline, W6, W14, M6, M9, M12} | Missing if no item answered |
| Social/family well-being subscore at Vi | 7 * (Sum of the items GS1 to GS7) / Number of items answered |
| Calculated for Vi = {Baseline, W6, W14, M6, M9, M12} | Missing if no item answered |
| Emotional well-being subscore at Vi | 6 * (Sum of the items GE1 to GE6) / Number of items answered |
| Calculated for Vi = {Baseline, W6, W14, M6, M9, M12} | Missing if no item answered |
| Functionnal well-being subscore at Vi | 7 * (Sum of the items GF1 to GF7) / Number of items answered |
| Calculated for Vi = {Baseline, W6, W14, M6, M9, M12} | Missing if no item answered |
| BMT subscore at Vi Calculated for Vi = {Baseline, W6, | 10 * (Sum of BMT1 to BMT4 + Sum of C6 to C7 + Sum of BMT5 to BMT6 + BL4 + BMT8) / Number of items answered |
| W14, M6, M9, M12} | Missing if no item answered |
| Global FACT-BMT score at Vi | The global FACT-BMT score is defined as the sum of all the subscores. |
| Calculated for Vi = {Baseine, W6, W14, M6, M9, M12} | Missing if at least one subscore is missing |
| Subscale score - Change from baseline at Vi | Subscale score at Vi – Subscale score at baseline |
| Calculated for Vi = {W6, W14, M6, M9, M12} and for physical well- | Missing if the subscore is missing at Vi and/or baseline |




| being, family/social well-being,<br>emotional well-being, functional well-<br>being and other concerns subscores | |
|---|---|
| Global FACT-BMT scale score -<br>Change from baseline at Vi | Global FACT-BMT score at Vi – Global FACT-BMT score at baseline |
| Calculated for Vi = {W6, W14, M6, M9, M12} | Missing if the global FACT-BMT is missing at Vi and/or baseline |

The following table will be presented:

| Variable | Visit | Statistics / Modality | FAS Population<br>(N = XX) |
|---|---|---|---|
| | | N (N Missing) | XX (XX) |
| | Baseline | Mean ± SD | $XX.X \pm XX.X$ |
| | Daseille | Median [Min ; Max] | XX [XX; XX] |
| | | CI 95% | (N = XX)<br>XX (XX)<br>XX.X ± XX.X |
| | | N (N Missing) | XX (XX) |
| | W6 | Mean ± SD | $XX.X \pm XX.X$ |
| | Median | Median [Min ; Max] | XX [XX; XX] |
| | | CI 95% | [XX.X; XX.X] |
| | | N (N Missing) | XX (XX) |
| | W14 | Mean ± SD | $XX.X \pm XX.X$ |
| | VV 1 <del>4</del> | Median [Min ; Max] | XX [XX; XX] |
| First subscore | | CI 95% | [XX.X; XX.X] |
| | MC | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | M6 | Median [Min ; Max] | XX [XX; XX] |
| | | CI 95% | [XX.X; XX.X] |
| | | N (N Missing) | XX (XX) |
| | M9 | Mean ± SD | $XX.X \pm XX.X$ |
| | IVI9 | Median [Min ; Max] | (N = XX) XX (XX) XX.X ± XX.X XX [XX; XX] [XX.X; XX.X] XX (XX) XX.X ± XX.X XX [XX; XX.] [XX.X; XX.X] XX (XX) XX.X ± XX.X XX [XX; XX.] [XX.X; XX.X] XX (XX) |
| | CI 95% | [XX.X; XX.X] | |
| | | N (N Missing) | XX (XX) |
| | N440 | Mean ± SD | $XX.X \pm XX.X$ |
| | M12 | Median [Min ; Max] | XX [XX; XX] |
| | | CI 95% | |
| First subsects Change | | N (N Missing) | XX (XX) |
| First subscore – Change | MG | Mean ± SD | |
| from baseline | W6 | Median [Min ; Max] | XX [XX; XX] |
| | | CI 95% | [XX.X; XX.X] |




| | N (N Missing) | XX (XX) |
|-------|--------------------|-----------------|
| W14 | Mean ± SD | $XX.X \pm XX.X$ |
| VV 14 | Median [Min ; Max] | XX [XX ; XX] |
| | CI 95% | [XX.X ; XX.X] |
| | N (N Missing) | XX (XX) |
| N40 | Mean ± SD | $XX.X \pm XX.X$ |
| M6 | Median [Min ; Max] | XX [XX ; XX] |
| | CI 95% | [XX.X ; XX.X] |
| | N (N Missing) | XX (XX) |
| 140 | Mean ± SD | $XX.X \pm XX.X$ |
| M9 | Median [Min ; Max] | XX [XX ; XX] |
| | CI 95% | [XX.X; XX.X] |
| | N (N Missing) | XX (XX) |
| MAO | Mean ± SD | $XX.X \pm XX.X$ |
| M12 | Median [Min ; Max] | XX [XX ; XX] |
| | CI 95% | [XX.X ; XX.X] |

This table will be completed for:

- Physical well-being subscore
- Social/family well-being subscore
- Emotional well-being subscore Eating and digestion subscore
- Functionnal subscore
- BMT subscore
- FACT-BMT score

Global score and each subscore over time will be graphically represented by boxplots.

The change from baseline over time of the global score and each subscore will be graphically represented by the mean and its associated CI 95%.

#### Lee Symptom Scale

#### **Derivation**

| Derived variables | Definition |
|---|---|
| Skin subscore at Vi | If at least 2 of the following items are answered, Scores are linearly transformed to a 0-100 scale where 0 |
| Calculated for Vi = {Baseline, W6, W14, M6, M9, M12} | means all answered items were a "0" and "100" means that all answered items were a "4" |
| , | |
| | Items: Abnormal skin color, Rashes, Thickened skin, Sores on skin and Itchy skin |



| | Missing otherwise |
|---|---|
| Eyes and mouth subscore at Vi Calculated for Vi = {Baseline, W6, W14, M6, M9, M12} | If at least 2 of the following items are answered, Scores are linearly transformed to a 0-100 scale where 0 means all answered items were a "0" and "100" means that all answered items were a "4" Items: Dry eyes, Need to use eyedrops frequently, Difficulty seeing clearly, Need to avoid certain foods due to mouth pain, Ulcers in mouth and Receiving nutrition from an intravenous line and feeding tube |
| | Missing otherwise |
| Breathing subscore at Vi Calculated for Vi = {Baseline, W6, W14, M6, M9, M12} | If at least 2 of the following items are answered, Scores are linearly transformed to a 0-100 scale where 0 means all answered items were a "0" and "100" means that all answered items were a "4" |
| | Items: Frequent cough, Colored sputum, Shortness of breath with exercise, Shortness of breath at rest and Need to use oxygen |
| | Missing otherwise |
| Eating and digestion subscore at Vi Calculated for Vi = {Baseline, W6, W14, M6, M9, M12} | If at least 2 of the following items are answered, Scores are linearly transformed to a 0-100 scale where 0 means all answered items were a "0" and "100" means that all answered items were a "4" |
| | Items: Difficulty swallowing solid foods, Difficulty swallowing liquids, Vomiting and Weight loss |
| | Missing otherwise |
| Muscles and joints subscore at Vi Calculated for Vi = {Baseline, W6, W14, M6, M9, M12} | If at least 2 of the following items are answered, Scores are linearly transformed to a 0-100 scale where 0 means all answered items were a "0" and "100" means that all answered items were a "4" |
| | Items: Joint and muscle aches, Limited joint movement, Muscle cramps and Weak muscles |
| | Missing otherwise |



| Energy subscore at Vi Calculated for Vi = {W6, W14, M6, M9, M12} | If at least 2 of the following items are answered, Scores are linearly transformed to a 0-100 scale where 0 means all answered items were a "0" and "100" means that all answered items were a "4" |
|---|---|
| | Items: Loss of energy, Need to sleep more/take naps and Fevers |
| | Missing otherwise |
| Mental and emotional subscore at Vi Calculated for Vi = {Baseline, W6, W14, M6, M9, M12} | If at least 2 of the following items are answered, Scores are linearly transformed to a 0-100 scale where 0 means all answered items were a "0" and "100" means that all answered items were a "4" |
| | Items: Depression, Anxiety and Difficulty sleeping |
| | Missing otherwise |
| Global Lee symptom scale score at Vi | The global score is defined as the average of subscores, if at least 4 are available. |
| Calculated for Vi = {Baseline, W6, W14, M6, M9, M12} | Missing otherwise |
| Subscale score - Change from baseline at Vi | Subscale score at Vi – Subscale score at baseline |
| Calculated for Vi = {W6, W14, M6, M9, M12} and for skin, eyes and mouth, breathing, eating and digestion, muscles and joints, energy, mental and emotional subscores | Missing if the subscore is missing at Vi and/or baseline |
| Global Lee symptom scale score -<br>Change from baseline at Vi | Global Lee score at Vi – Global Lee score at baseline |
| Calculated for Vi = {W6, W14, M6, M9, M12} | Missing if the global Lee score is missing at Vi and/or baseline |




## The following table will be presented:

| Variable | Visit | Statistics / Modality | FAS Population<br>(N = XX) |
|---|---|---|---|
| | | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | Baseline | Median [Min ; Max] | XX [XX ; XX] |
| | | CI 95% | [XX.X; XX.X] |
| | | N (N Missing) | XX (XX) |
| | W6 | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX ; XX] |
| | | CI 95% | [XX.X ; XX.X] |
| | | N (N Missing) | XX (XX) |
| | W14 | Mean ± SD | XX.X ± XX.X |
| First subscore | | Median [Min ; Max] | XX [XX ; XX] |
| 1 1101 00000010 | - | CI 95% | [XX.X ; XX.X] |
| | | N (N Missing) | XX (XX) |
| | M6 | Mean ± SD | $XX.X \pm XX.X$ |
| | • | Median [Min ; Max] | XX [XX ; XX] |
| | | CI 95% | [XX.X ; XX.X] |
| | | N (N Missing) | XX (XX) |
| | M9 | Mean ± SD | $XX.X \pm XX.X$ |
| | 1110 | Median [Min ; Max] | XX [XX ; XX] |
| | | CI 95% | [XX.X ; XX.X] |
| | | N (N Missing) | XX (XX) |
| | M12 | Mean ± SD | $XX.X \pm XX.X$ |
| | IVI I Z | Median [Min ; Max] | XX [XX ; XX] |
| | | CI 95% | [XX.X; XX.X] |
| | | N (N Missing) | XX (XX) |
| | W6 | Mean ± SD | $XX.X \pm XX.X$ |
| | **** | Median [Min ; Max] | XX [XX; XX] |
| | | CI 95% | [XX.X ; XX.X] |
| | | N (N Missing) | XX (XX) |
| | W14 | Mean ± SD | $XX.X \pm XX.X$ |
| First subscore – Change | ** 1 1 | Median [Min ; Max] | XX [XX ; XX] |
| from baseline | - | CI 95% | [XX.X; XX.X] |
| | | N (N Missing) | XX (XX) |
| | M6 | Mean ± SD | $XX.X \pm XX.X$ |
| | IVIO | Median [Min ; Max] | XX [XX; XX] |
| | - | CI 95% | [XX.X ; XX.X] |
| | | N (N Missing) | XX (XX) |
| | M9 | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX; XX] |




| | CI 95% | [XX.X ; XX.X] |
|---------|--------------------|-----------------|
| | N (N Missing) | XX (XX) |
| M12 | Mean ± SD | $XX.X \pm XX.X$ |
| IVI I Z | Median [Min ; Max] | XX [XX; XX] |
| | CI 95% | [XX.X ; XX.X] |

This table will be completed for:

- Skin subscore
- Eyes and mouth subscore
- Breathing subscore
- Eating and digestion subscore
- Energy subscore
- Mental and emotional subscore
- Global Lee symptom scale score

Global score and each subscore over time will be graphically represented by boxplots.

The change from baseline over time of the global score and each subscore will be graphically represented by the mean and its associated CI 95%.

## 11.4.2.5 Assessment of chronic GvHD activity post-ATO treatment

Chronic GvHD activity (global and by organ) will be reported at 6 weeks, 14 weeks, 6, 9 and 12 months after the first infusion of ATO.

#### Global chronic GvHD activity

| Variable | Modality | FAS Population<br>(N = XX) |
|------------------------|---------------|----------------------------|
| Health care provider g | lobal ratings | |
| W6 | None | n/N (XX.XX%) |
| | Mild | n/N (XX.XX%) |
| | Moderate | n/N (XX.XX%) |
| | Severe | n/N (XX.XX%) |
| | Missing | n |
| W14 | None | n/N (XX.XX%) |
| | Mild | n/N (XX.XX%) |
| | Moderate | n/N (XX.XX%) |
| | Severe | n/N (XX.XX%) |




| | Missing | n |
|-----|----------|--------------|
| M6 | None | n/N (XX.XX%) |
| | Mild | n/N (XX.XX%) |
| | Moderate | n/N (XX.XX%) |
| | Severe | n/N (XX.XX%) |
| | Missing | n |
| M9 | None | n/N (XX.XX%) |
| | Mild | n/N (XX.XX%) |
| | Moderate | n/N (XX.XX%) |
| | Severe | n/N (XX.XX%) |
| | Missing | n |
| M12 | None | n/N (XX.XX%) |
| | Mild | n/N (XX.XX%) |
| | Moderate | n/N (XX.XX%) |
| | Severe | n/N (XX.XX%) |
| | Missing | 'n |

Stacked bar graphs will be used for illustrating the percentage of patients in each score category at each time points (6 weeks, 14 weeks, 6, 9 and 12 months after the first infusion of ATO).

#### • Chronic GvHD activity for each organ

#### o **Derivation**

| Derived variables | Definition |
|---|---|
| Mouth score | For each visit of interest, sum of the 3 following scores: |
| | - Erythema (MOUTH1) |
| | - Lichenoid (MOUTH2) |
| | - Ulcers (MOUTH3) |
| | Missing if at least one missing score |
| | Score to be calculated for the following visits: W6, W14, M6, M9 and M12 |




The following table will be presented:

| 0 | \/:~!4 | Otatiatias / Madality | FAS Population<br>(N=XX) |
|---|---|---|---|
| Organ score | Visit | Statistics / Modality | |
| Organ – Abnormalities | W6 | No | n/N (XX.X%) |
| present but explained entirely by non-GvHD documented | | Yes | n/N (XX.X%) |
| cause | | Missing | n |
| Categorical score | W6 | Modality 1 | n/N (XX.XX%) |
| | | Modality n | n/N (XX.XX%) |
| | | Missing | n |
| Organ – Abnormalities | W14 | No | n/N (XX.X%) |
| present but explained entirely | | Yes | n/N (XX.X%) |
| oy non-GvHD documented cause | | Missing | n |
| Categorical score | W14 | Modality 1 | n/N (XX.XX%) |
| | | Modality n<br>Missing | n/N (XX.XX%)<br>n |
| Organ – Abnormalities | M6 | No | n/N (XX.X%) |
| present but explained entirely | | Yes | n/N (XX.X%) |
| by non-GvHD documented cause | | Missing | n |
| Categorical score | M6 | Modality 1 | n/N (XX.XX%) |
| | | <br>Modality n | n/N (XX.XX%) |
| | | Missing | n |
| Organ – Abnormalities | M9 | No | n/N (XX.X%) |
| present but explained entirely | | Yes | n/N (XX.X%) |
| | | Missing | n |




# by non-GvHD documented cause

| Categorical score | M9 | Modality 1 | n/N (XX.XX%) |
|--------------------------------|-----|--------------------|------------------|
| | | <br>Modality n | <br>n/N (XX.XX%) |
| | | Missing | n |
| Organ – Abnormalities | M12 | No | n/N (XX.X%) |
| present but explained entirely | | Yes | n/N (XX.X%) |
| by non-GvHD documented | | | ( |
| cause | | Missing | n |
| Categorical score | M12 | Modality 1 | n/N (XX.XX%) |
| | | <br>Modality n | n/N (XX.XX%) |
| | | Missing | ` n |
| Liver – Abnormalities present | W6 | No | n/N (XX.X%) |
| but explained entirely by non- | | Yes | n/N (XX.X%) |
| GvHD documented cause | | 103 | 11/14 (703.7570) |
| | | Missing | n |
| Total bilirubin* | W6 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX; XX] |
| SGPT* | W6 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX; XX] |
| ALK* | W6 | N (N Missing) | XX (XX) |
| | | Mean ± SD | XX.X ± XX.X |
| | | Median [Min ; Max] | XX [XX; XX] |
| Lung – Abnormalities present | W6 | No | n/N (XX.X%) |
| but explained entirely by non- | | Yes | n/N (XX.X%) |
| GvHD documented cause | | 1.00 | 1111 (700.7070) |
| | | Missing | n |
| FEV1** | W6 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |



| | | Median [Min ; Max] | XX [XX ; XX] |
|---|---|---|---|
| Liver – Abnormalities present | W14 | No | n/N (XX.X%) |
| but explained entirely by non- | | Yes | n/N (XX.X%) |
| GvHD documented cause | | 165 | 11/IN (AA.A70) |
| CVID GOGGINGING GGGG | | Missing | n |
| Total bilirubin* | W14 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX ; XX] |
| SGPT* | W14 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX ; XX] |
| ALK* | W14 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | 11111 | Median [Min ; Max] | XX [XX ; XX] |
| Lung – Abnormalities present | W14 | No | n/N (XX.X%) |
| but explained entirely by non- | | Yes | n/N (XX.X%) |
| GvHD documented cause | | | () |
| | | Missing | n |
| FEV1** | W14 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX ; XX] |
| Liver – Abnormalities present | M6 | No | n/N (XX.X%) |
| but explained entirely by non- | | Yes | n/N (XX.X%) |
| GvHD documented cause | | 100 | 11/14 (703.7470) |
| | | Missing | n |
| Total bilirubin* | M6 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX; XX] |
| SGPT* | M6 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX ; XX] |
| ALK* | M6 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX ; XX] |
| Lung – Abnormalities present | M6 | No | n/N (XX.X%) |
| but explained entirely by non- | | Yes | n/N (XX.X%) |
| GvHD documented cause | | . •• | (- 5 ) |
| | | Missing | n |
| FEV1** | M6 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX ; XX] |



| Liver – Abnormalities present | M9 | No | n/N (XX.X%) |
|---|---|---|---|
| but explained entirely by non- | | Vaa | ~/NI /VV V0/ ) |
| GvHD documented cause | | Yes | n/N (XX.X%) |
| CVI D documented cause | | Missing | n |
| Total bilirubin* | M9 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX ; XX] |
| SGPT* | M9 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX ; XX] |
| ALK* | M9 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX ; XX] |
| Lung – Abnormalities present | M9 | No | n/N (XX.X%) |
| but explained entirely by non- | | Yes | n/N /VV V0/.) |
| GvHD documented cause | | 165 | n/N (XX.X%) |
| OVI ID documented cause | | Missing | n |
| FEV1** | M9 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX; XX] |
| Liver – Abnormalities present | M12 | No | n/N (XX.X%) |
| but explained entirely by non- | | Yes | n/N (XX.X%) |
| GvHD documented cause | | 100 | 11/14 (704.7470) |
| | | Missing | n |
| Total bilirubin* | M12 | N (N Missing) | XX (XX) |
| | | Mean ± SD | XX.X ± XX.X |
| | | Median [Min ; Max] | XX [XX ; XX] |
| SGPT* | M12 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX ; XX] |
| ALK* | M12 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX ; XX] |
| Lung – Abnormalities present | M12 | No | n/N (XX.X%) |
| but explained entirely by non- | | Yes | n/N (XX.X%) |
| GvHD documented cause | | | (/-) |
| | | Missing | n |
| FEV1** | M12 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| * Chamistry apposited to liver ** | | Median [Min ; Max] | XX [XX ; XX] |

<sup>\*</sup> Chemistry associated to liver, \*\* Linked to lung function




## This table will be completed for the following scores:

| Organ | Score |
|---|---|
| Skin | Score 0: No BSA involved |
| | Score 1: 1-18% BSA |
| | Score 2: 19-50% BSA<br>Score 3: > 50% BSA |
| Skin features score | Score 0: No sclerotic features |
| Skill leatures score | Score of No scierotic leatures |
| | Score 2: Superficial sclerotic features "not |
| | hidebound" (able to pinch) |
| | , , , |
| | Score 3: Deep sclerotic features, |
| | "Hidebound" (unable to pinch), Impaired |
| | mobility, Ulceration |
| Mouth Enthoma | None |
| Mouth - Erythema | Mild erythema or moderate erythema |
| | (<25%) |
| | Moderate (>=25%) or severe erythema |
| | (<25%) |
| | Severe erythema (>= 25%) |
| Mouth - Lichenoid | None |
| | Lichen-like changes (<25%) |
| | Lichen-like changes (25-50%) |
| Mouth - Ulcers | Lichen-like changes (>50%) |
| Mouth - Oicers | None Ulcers involving (<=20%) |
| | Severe ulcerations (>20%) |
| Eyes | Score 0: No symptoms |
| 2,00 | Coole of the cymptoms |
| | Score 1: Mild dry eye symptoms not |
| | affecting ADL |
| | Score 2: Moderate dry eye symptoms |
| | partially affecting ADL without new vision |
| | impairment due to KCS |
| | Score 3: Severe eye symptoms |
| | significantly affecting ADL or unable to |
| | work because of ocular symptoms of loss |
| | or vision due to KCS |
| Gastro-intestinal (Esophageal) | 0 = No esophageal symptoms |



| | 1 = Occasional dysphagia or odynophagia with solid foods or pills during the past week 2 = Intermittent dysphagia or odynophagia with solid foods or pills, but not for liquids or soft foods, during the past week 3 = Dysphagia or odynophagia for almost |
|---|---|
| | all oral intake, on almost every day of the past week |
| Gastro-intestinal (Upper) | 0 = No symptoms |
| | 1 = Mild, occasional symptoms, with little reduction in oral intake during the past week |
| | 2 = Moderate, intermittent symptoms, with some reduction in oral intake during the past week |
| | 3 = More severe or persistent symptoms throughout the day, with marked reduction in oral intake, on almost every day of the past week |
| Gastro-intestinal (Lower) | 0 = No loose or liquid stools during the past week |
| | 1 = Occasional loose or liquid stools, on some days during the past week |
| | 2 = Intermittent loose or liquid stools<br>throughout the day, on almost every day of<br>the past week, without requiring<br>intervention to prevent or correct volume<br>depletion |
| | 3 = Voluminous diarrhea on almost every day of the past week, requiring intervention to prevent or correct volume depletion |
| Joint and fascia | Score 0: No symptoms |




| | Score 1: Mild tightness of arms or legs,<br>normal or mild decreased range of motion<br>and not affecting ADL |
|---|---|
| | Score 2: Tightness of arms or legs OR joint contractures, erythema thought due to fasciitis, moderate decrease ROM AND mild to moderate limitation of ADL |
| | Score 3 : Contractures WITH significant decrease |
| | of ROM AND significant limitation of ADL (unable to tie shoes, button shirts, dress self, etc.) |
| Lungs | Score 0: No symptoms |
| | Score 1: Mild symptoms (shortness or breath after climbing one flight of steps) |
| | Score 2: Moderate symptoms (shortness of breath after walking on flat ground) |
| | Score 3: Severe symptoms (shortness of breath at rest, requiring O2) |

This table will be also presented on PP population.

Stacked bar graphs will be used for illustrating the percentage of patients in each score category at each time points (6 weeks, 14 weeks, 6, 9 and 12 months after the first infusion of ATO).

Continuous indicators will be represented by boxplots.

#### • Physician assessment of current overall chronic GvHD severity

| Variable | Statistics | FAS Population<br>(N = XX) |
|---|---|---|
| Chronic GVHD seve | erity from 0 (not at all) to 10 (the m | ost severe) |
| W6 | N (N Missing) | XX (XX) |
| | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| W14 | N (N Missing) | XX (XX) |
| | Mean ± SD | $XX.X \pm XX.X$ |




| | Median [Min ; Max] | XX [XX ; XX] |
|-----|--------------------|-----------------|
| M6 | N (N Missing) | XX (XX) |
| | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX; XX] |
| M9 | N (N Missing) | XX (XX) |
| | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX; XX] |
| M12 | N (N Missing) | XX (XX) |
| | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |

Physician evaluations of current overall chronic GvHD severity over time will be graphically represented by boxplots.

## • Physician evaluations of chronic GvHD changes

| Variable | Statistics | FAS Population<br>(N = XX) |
|---|---|---|
| Over the time would ye | ou say that this patient's GVHD | is |
| W6 | N (N Missing) | XX (XX) |
| | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |
| W14 | N (N Missing) | XX (XX) |
| | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX; XX] |
| M6 | N (N Missing) | XX (XX) |
| | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX; XX] |
| M9 | N (N Missing) | XX (XX) |
| | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX; XX] |
| M12 | N (N Missing) | XX (XX) |
| | Mean ± SD | $XX.X \pm XX.X$ |
| | Median [Min ; Max] | XX [XX ; XX] |

Physician evaluations of chronic GvHD changes over time will be graphically represented by boxplots.




#### 12. SAFETY EVALUATION

#### 12.1 ADVERSE EVENTS

All treatment related toxicities and other AE and SAE occurring from the time of signed informed consent until the end of the study are recorded. They are coded using the Medical Dictionary for Regulatory Activities (MedDRA) and classified according to the NCI common toxicity criteria (CTC), specification for stem cell transplantation.

A SAE or serious adverse drug reaction is any untoward medical occurrence at any dose that:

- Results in death;
- Is life-threatening (immediate risk of death);
- Requires inpatient hospitalization or prolongation of existing hospitalization for medical reasons (e.g. prolongation of hospitalization for social reasons is excluded):
- · Results in persistent or significant disability/incapacity;
- Results in congenital anomaly/birth defect.

The investigator will decide whether the serious adverse event is related to trial medication. The decision will be recorded on the serious adverse event report.

The assessment of causality is made by the investigator as not related, unlikely, possibly related or definitely related.

All AE not previously described in the Summary of Product Characteristics of TRISENOX® or in the Investigator Brochure of ARSCIMED® should be considered as unexpected AE.

When calculating the incidence of AEs and SAEs, each subject will only be counted once and any repetitions of AEs will be ignored; the denominator will be the total population size.




| Type of AE | Safety Population<br>(N=XX) | N AEs |
|--------------------------|-----------------------------|-------|
| AE | n/N (XX.X%) | n |
| Serious AE | n/N (XX.X%) | n |
| AE leading to death | n/N (XX.X%) | n |
| AE leading to withdrawal | n/N (XX.X%) | n |
| Related AE | n/N (XX.X%) | n |

Adverse events will be also presented by SOC and PT:

| soc | PT | Safety Population (N=XX) | N AEs |
|-------|------|--------------------------|-------|
| | PT 1 | n/N (XX.X%) | n |
| SOC 1 | PT 2 | n/N (XX.X%) | n |
| | PT 1 | n/N (XX.X%) | n |
| SOC n | PT 2 | n/N (XX.X%) | n |

This table will be presented for each type of AE.

A list of all AEs will be produced in a table including the following items:

- Patient number
- Age at inclusion
- AE names
- AE grade
- Seriousness
- Date of onset first cycle ATO
- Date of end first cycle ATO
- Second cycle ATO (yes/no)
- Date of onset second cycle ATO
- Date of end second cycle ATO




- Relation (causality)
- Action taken for AE
- Date of onset of AE
- Outcome of AE (Resolved without sequelae/ ongoing/ death)

#### 12.2 LABORATORY PARAMETERS

Each laboratory parameter will be described at baseline, W6, W14, M6, M9 and M12 and presented as follows:

| Variable | Visit | Statistics / Modality | Safety Population<br>(N = XX) |
|---|---|---|---|
| | | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | Dagalina | Median [Min ; Max] | XX [XX; XX] |
| | Baseline | Not clinically significant | n/N (XX.X%) |
| | | Clinically significant | n/N (XX.X%) |
| | | Missing | n |
| | | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | 14/0 | Median [Min ; Max] | XX [XX; XX] |
| | W6 | Not clinically significant | n/N (XX.X%) |
| | | Clinically significant | n/N (XX.X%) |
| | | Missing | n |
| aboratory parameter 1 | W14 | N (N Missing) | XX (XX) |
| aboratory parameter | | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX; XX] |
| | | Not clinically significant | n/N (XX.X%) |
| | | Clinically significant | n/N (XX.X%) |
| | | Missing | n |
| | | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| | MC | Median [Min ; Max] | XX [XX; XX] |
| | M6 | Not clinically significant | n/N (XX.X%) |
| | | Clinically significant | n/N (XX.X%) |
| | | Missing | n |
| | | N (N Missing) | XX (XX) |
| | M9 | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX; XX] |




| | Not clinically significant<br>Clinically significant<br>Missing | n/N (XX.X%)<br>n/N (XX.X%)<br>n |
|---|---|---|
| | N (N Missing)<br>Mean ± SD<br>Median [Min ; Max] | XX (XX)<br>XX.X ± XX.X<br>XX [XX ; XX] |
| M12 | Not clinically significant<br>Clinically significant<br>Missing | n/N (XX.X%)<br>n/N (XX.X%)<br>n |

. . .

This table will be completed for the following parameters:

- Leucocytes
- Neutrophils
- Lymphocytes
- Monocytes
- Eosinophils
- Hemoglobin
- Platelets
- PR
- aPTT
- Glycaemia
- Creatinine
- Uric acid
- Calcium
- Potassium
- Magnesium
- Total protein




- Albumin
- Total bilirubin
- Alkaline phosphatases
- SGOT (ASAT)
- SGPT (ALAT)
- LDH

#### 12.3 PHYSICAL EXAMINATION

Each body system of the clinical examination will be described at baseline, W6, W14, M6, M9 and M12 and presented as follows:

| Variable | Visit | Statistics | Safety Population<br>(N = XX) |
|-------------|----------|--------------------|-------------------------------|
| | | N (N Missing) | XX (XX) |
| | Baseline | Mean ± SD | $XX.X \pm XX.X$ |
| | Daseille | Median [Min ; Max] | XX [XX; XX] |
| | | N (N Missing) | XX (XX) |
| | W6 | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX; XX] |
| | W14 | N (N Missing) | XX (XX) |
| | | Mean ± SD | $XX.X \pm XX.X$ |
| Parameter 1 | | Median [Min ; Max] | XX [XX; XX] |
| | | N (N Missing) | XX (XX) |
| | M6 | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX; XX] |
| | | N (N Missing) | XX (XX) |
| | M9 | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX; XX] |
| | | N (N Missing) | XX (XX) |
| | M12 | Mean ± SD | $XX.X \pm XX.X$ |
| | | Median [Min ; Max] | XX [XX; XX] |

. . .




## This table will be completed for the following parameters:

- Cardiac frequency
- Systolic arterial pressure
- Diastolic arterial pressure
- Temperature
- O2 saturation




#### 13. DISCUSSION AND OVERALL CONCLUSIONS

At the end of the study evaluation, the principle investigator presents a final report, containing the clinical report, single tables, and the final conclusions. Publication of the results is realized independently from the outcome of the study. The study or parts of the study should be published by the writing committee only which consists of the persons in charge of the study as mentioned on the front page. According to the EBMT rules, coauthors will be offered to the local PI of participating centres, the order depending on the number of patients included by the respective centres, or depending on their contribution to the protocol or the realization of the study. Other investigators will be mentioned in the addendum. All publications and/or communications related to this study should at least mention the PI of the study and the sponsor.




#### 14. TABLES, FIGURES AND GRAPHS

## **14.1 TABLES**

| Table<br>Number | Population | Table Title / Summary |
|---|---|---|
| 14.1 Demog | raphic and Baselin | e Data |
| | sition and Deviation | |
| 14.1.1.1 | All Patients | Study Disposition |
| 14.1.1.2 | All Patients | Protocol Deviations |
| 14.1.1.3 | All Patients | Analyses Populations |
| 14.1.2 Demo | graphic Data and | other baseline characteristics |
| 14.1.2.1 | Safety | Demographic characteristics |
| 14.1.2.2 | Safety | Baseline characteristics |
| 14.1.2.3 | Safety | Signs and symptoms of cGvHD at baseline |
| 14.1.3 ATO | and associated trea | |
| 14.1.3.1 | Safety | Arsenic trioxide therapy |
| 14.1.4.1 | Safety | Associated treatment |
| 14.1.4.2 | Safety | Concomitant treatments |
| 14.1.4.3 | Safety | Secondary immunosuppressive treatment |
| 14.2 Efficac | y – Primary criterio | on Control of the Con |
| 14.2.1 Main | analyses | |
| 14.2.1.1 | FAS | Complete or partial response at 6 months (PI response) – Overall |
| 14.2.1.2 | FAS | Complete and partial response at 6 months (PI response) – Overall |
| 14.2.1.3 | FAS | Complete or partial response at 6 months (PI response) – By sex |
| 14.2.1.4 | FAS | Complete and partial response at 6 months (PI response) – By sex |
| 14.2.1.5 | FAS | Complete or partial response at 6 months (PI response) – By center |
| 14.2.1.6 | FAS | Complete and partial response at 6 months (PI response) – By center |
| 14.2.1.7 | FAS | Complete or partial response at 6 months (PI response) – By number of cycles of ATO |
| 14.2.1.8 | FAS | Complete and partial response at 6 months (PI response) – By number of cycles of ATO |
| 14.2.1.9 | FAS | Complete or partial response at 6 months (PI response) – By use of Ciclosporin or not |
| 14.2.1.10 | FAS | Complete and partial response at 6 months (PI response) – By use of Ciclosporin or not |
| 14.2.1.11 | FAS | Complete or partial response at 6 months (PI response) – By number of organs involved in cGvHD |



| Table<br>Number | Population | Table Title / Summary |
|---|---|---|
| 14.2.1.12 | FAS | Complete and partial response at 6 months (PI response) – By number of organs involved in cGvHD |
| 14.2.1.13 | FAS | Complete or partial response at 6 months (PI response) – By GvHD severity at baseline |
| 14.2.1.14 | FAS | Complete and partial response at 6 months (PI response) – By GvHD severity at baseline |
| 14.2.2 Sensi | tivity analyses | |
| 14.2.2.1 | PP | Complete or partial response at 6 months (PI response) – Overall |
| 14.2.2.2 | PP | Complete and partial response at 6 months (PI response) – Overall |
| 14.2.2.3 | FAS | Complete or partial response at 6 months (computed response) – Overall |
| 14.2.2.4 | FAS | Complete and partial response at 6 months (computed response) – Overall |
| 14.2.2.5 | FAS | Complete or partial response at 6 months (computed response) – By sex |
| 14.2.2.6 | FAS | Complete and partial response at 6 months (computed response) – By sex |
| 14.2.2.7 | FAS | Complete or partial response at 6 months (computed response) – By center |
| 14.2.2.8 | FAS | Complete and partial response at 6 months (computed response) – By center |
| 14.2.2.9 | FAS | Complete or partial response at 6 months (computed response) – By number of cycles of ATO |
| 14.2.2.10 | FAS | Complete and partial response at 6 months (computed response) – By number of cycles of ATO |
| 14.2.2.11 | FAS | Complete or partial response at 6 months (computed response) – By use of Ciclosporin or not |
| 14.2.2.12 | FAS | Complete and partial response at 6 months (computed response) – By use of Ciclosporin or not |
| 14.2.2.13 | FAS | Complete or partial response at 6 months (computed response) – By number of organs involved in cGvHD |
| 14.2.2.14 | FAS | Complete and partial response at 6 months (computed response) – By number of organs involved in cGvHD |
| 14.2.2.15 | FAS | Complete or partial response at 6 months (computed response) – By GvHD severity at baseline |
| 14.2.2.16 | FAS | Complete and partial response at 6 months (computed response) – By GvHD severity at baseline |
| 14.2.2.17 | FAS | Complete or partial response at 6 months (PI response) without patients 06-07, 06-08 and 06-09 — Overall |
| 14.2.2.18 | FAS | Complete and partial response at 6 months (PI response) without patients 06-07, 06-08 and 06-09 — Overall |
| 14.2.2.19 | FAS | Complete or partial response at 6 months (computed response) without patients 06-07, 06-08 and 06-09 — Overall |



| Table<br>Number | Population | Table Title / Summary |
|---|---|---|
| 14.2.2.20 | FAS | Complete and partial response at 6 months (computed response) without patients 06-07, 06-08 and 06-09 – Overall |
| 14.3 Efficacy | - Secondary crite | eria |
| 14.3.1 Respo | onse at 6 months b | oy organ |
| 14.3.1 | FAS | Response at 6 months by organ |
| 14.3.2 | PP | Response at 6 months by organ |
| 14.3.2 Surviv | al analyses | |
| 14.3.2.1a | FAS | Failure free survival at M6 |
| 14.3.2.1B | PP | Failure free survival at M6 |
| 14.3.2.2a | FAS | Failure free survival at M12 |
| 14.3.2.2b | PP | Failure free survival at M12 |
| 14.3.2.3a | FAS | Progression free survival at M6 |
| 14.3.2.3b | PP | Progression free survival at M6 |
| 14.3.2.4a | FAS | Progression free survival at M12 |
| 14.3.2.4b | PP | Progression free survival at M12 |
| 14.3.2.5a | FAS | Overall survival at M6 |
| 14.3.2.5b | PP | Overall survival at M6 |
| 14.3.2.6a | FAS | Overall survival at M12 |
| 14.3.2.6b | PP | Overall survival at M12 |
| 14.3.3 Treatn | nent by corticoste | roids |
| 14.3.3.1 | FAS | Treatment by corticosteroids by visit – Absolute values and change from baseline |
| 14.3.4 Qualit | 14.3.4 Quality of life assessment | |
| 14.3.4.1 | FAS | FACT-BMT by visit – Absolute values and change from baseline |
| 14.3.4.2 | FAS | Lee symptom scale by visit – Absolute values and change from baseline |
| 14.3.5 Asses | sment of chronic | GVHD activity post-ATO treatment |
| 14.3.5.1 | FAS | Global chronic GVHD activity by visit |




| Table<br>Number | Population | Table Title / Summary |
|---|---|---|
| 14.3.5.2 | FAS | Chronic GVHD activity for each organ by visit |
| 14.3.5.3 | FAS | Physician assessment of current overall chronic GVHD severity by visit |
| 14.3.5.4 | FAS | Physician evaluations of chronic GVHD changes by visit |
| 14.4 Safety | • | |
| 14.4.1 Advers | se events | |
| 14.4.1.1 | Safety | AEs summary – During treatment (Cycle 1 and/or Cycle 2) |
| 14.4.1.2 | Safety | AEs summary - After the last infusion of ATO until 6 months after the first infusion of ATO |
| 14.4.1.3 | Safety | AEs summary - From 6 to 12 months after the first infusion of ATO |
| 14.4.1.4 | Safety | AEs by SOC/PT |
| 14.4.1.5 | Safety | SAEs by SOC/PT |
| 14.4.1.6 | Safety | AEs leading to death by SOC/PT |
| 14.4.1.7 | Safety | AEs leading to withdrawal by SOC/PT |
| 14.4.1.8 | Safety | Related AEs by SOC/PT |
| 14.4.2: Labor | ratory parameters | 1 |
| 14.4.2.1 | Safety | Laboratory parameters by visit – Absolute values |
| 14.4.3: Physi | cal examination | <u>'</u> |
| 14.4.3.1 | Safety | Physical examination by visit – Absolute values |

## 14.2 FIGURES AND GRAPHS

| Figure<br>Number | Population | Figure Title / Summary |
|---|---|---|
| 14.2 Efficacy | 14.2 Efficacy – Primary criterion | |
| 14.2.1 Main a | 14.2.1 Main analyses | |
| 14.2.1.1 | FAS | Forest plot of Complete and partial response at 6 months (PI response) |
| 14.2.2 Sensit | 14.2.2 Sensitivity analyses | |
| 14.2.2.1 | PP | Forest plot of Complete and partial response at 6 months (PI response) |



| 44000 | 1540 | |
|---|---|---|
| 14.2.2.2 | FAS | Forest plot of Complete and partial response at 6 months (computed response) |
| 14.2.2.3 | FAS | Forest plot of Complete and partial response at 6 months (PI response) without patients 06-07, 06-08 and 06-09 |
| 14.2.2.4 | FAS | Forest plot of Complete and partial response at 6 months (computed response) without patients 06-07, 06-08 and 06-09 |
| 14.3 Efficacy | - Secondary crit | |
| 14.3.1 Surviv | al analyses | |
| 14.3.1.1a | FAS | Kaplan-Meier survival plot of Failure free survival at M6 |
| 14.3.1.1b | PP | Kaplan-Meier survival plot of Failure free survival at M6 |
| 14.3.1.2a | FAS | Kaplan-Meier survival plot of Failure free survival at M12 |
| 14.3.1.2b | PP | Kaplan-Meier survival plot of Failure free survival at M12 |
| 14.3.1.3a | FAS | Kaplan-Meier survival plot of Progression free survival at M6 |
| 14.3.1.3b | PP | Kaplan-Meier survival plot of Progression free survival at M6 |
| 14.3.1.4a | FAS | Kaplan-Meier survival plot of Progression free survival at M12 |
| 14.3.1.4b | PP | Kaplan-Meier survival plot of Progression free survival at M12 |
| 14.3.1.5a | FAS | Kaplan-Meier survival plot of Overall survival at M6 |
| 14.3.1.5b | PP | Kaplan-Meier survival plot of Overall survival at M6 |
| 14.3.1.6a | FAS | Kaplan-Meier survival plot of Overall survival at M12 |
| 14.3.1.6b | PP | Kaplan-Meier survival plot of Overall survival at M12 |
| 14.3.2 Treatr | nent by corticoste | eroids |
| 14.3.2.1 | FAS | Stacked bars of Prednisone dose by visit |
| 14.3.2.2 | FAS | Stacked bars of change from baseline of Prednisone dose by visit |
| 14.3.3 Qualit | y of life assessme | ent |
| 14.3.3.1.1a | FAS | Boxplot of FACT-BMT Physical well-being subscore by visit |
| 14.3.3.1.1b | FAS | Boxplot of change from baseline of FACT-BMT Physical well-being subscore by visit |
| 14.3.3.1.2a | FAS | Boxplot of FACT-BMT Social/Family well-being subscore by visit |
| 14.3.3.1.2b | FAS | Boxplot of change from baseline of FACT-BMT Social/Family well-being subscore by visit |



| 14.3.3.1.3a | FAS | Boxplot of FACT-BMT Emotional subscore by visit |
|---|---|---|
| 14.3.3.1.3b | FAS | Boxplot of change from baseline of FACT-BMT Emotional well-<br>being subscore by visit |
| 14.3.3.1.4a | FAS | Boxplot of FACT-BMT Functionnal subscore by visit |
| 14.3.3.1.4b | FAS | Boxplot of change from baseline of FACT-BMT Functionnal subscore by visit |
| 14.3.3.1.5a | FAS | Boxplot of FACT-BMT Other concerns subscore by visit |
| 14.3.3.1.5b | FAS | Boxplot of change from baseline of FACT-BMT Other concerns subscore by visit |
| 14.3.3.1.6a | FAS | Boxplot of global FACT-BMT score by visit |
| 14.3.3.1.6b | FAS | Boxplot of change from baseline of global FACT-BMT score by visit |
| 14.3.3.2.1a | FAS | Boxplot of Lee symptom scale skin subscore by visit |
| 14.3.3.2.1b | FAS | Boxplot of change from baseline of Lee symptom scale skin subscore by visit |
| 14.3.3.2.2a | FAS | Boxplot of Lee symptom scale eyes and mouth subscore by visit |
| 14.3.3.2.2b | FAS | Boxplot of change from baseline of Lee symptom scale eyes and mouth subscore by visit |
| 14.3.3.2.3a | FAS | Boxplot of Lee symptom scale breathing subscore by visit |
| 14.3.3.2.3b | FAS | Boxplot of change from baseline of Lee symptom scale breathing subscore by visit |
| 14.3.3.2.4a | FAS | Boxplot of Lee symptom scale eating and digestion subscore by visit |
| 14.3.3.2.4b | FAS | Boxplot of change from baseline of Lee symptom scale eating and digestion subscore by visit |
| 14.3.3.2.5a | FAS | Boxplot of Lee symptom scale energy subscore by visit |
| 14.3.3.2.5b | FAS | Boxplot of change from baseline of Lee symptom scale energy subscore by visit |
| 14.3.3.2.6a | FAS | Boxplot of Lee symptom scale mental and emotional subscore by visit |
| 14.3.3.2.6b | FAS | Boxplot of change from baseline of Lee symptom scale mental and emotional subscore by visit |
| 14.3.3.2.7a | FAS | Boxplot of Global Lee symptom scale subscore by visit |
| 14.3.3.2.7b | FAS | Boxplot of change from baseline of Global Lee symptom scale subscore by visit |
| 14.3.4 Asses | sment of chronic | GVHD activity post-ATO treatment |
| 14.3.4.1 | FAS | Stacked bars of Global chronic GVHD activity by visit |



| 14.3.4.2 | FAS | Stacked bars of Chronic GVHD activity for each organ by visit |
|---|---|---|
| 14.3.4.3 | FAS | Boxplot of total bilirubin by visit |
| 14.3.4.4 | FAS | Boxplot of ALT (SGPT) by visit |
| 14.3.4.5 | FAS | Boxplot of PAL (ALK) by visit |
| 14.3.4.6 | FAS | Boxplot of FEV1 by visit |
| 14.3.4.7 | FAS | Boxplots of Physician assessment of current overall chronic GVHD severity by visit |
| 14.3.4.8 | FAS | Boxplots of Physician evaluations of chronic GVHD changes by visit |



### 15. REFERENCE LIST

A'Hern R.P. Sample size tables for exact single-stage phase II designs. Statistics in

Medicine. 2001; 20: 859-866).

Gamble C et al. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials JAMA December 19, 2017 Volume 318, Number 23




## 16. LISTINGS

| Listing<br>Number | Listing Title / Summary |
|---|---|
| 16.2.1 Discontinued patients | |
| 16.2.1.1 | Study Completion |
| 16.2.1.2 | Visits and Dates of Visits |
| 16.2.2 Protoc | ol Deviations |
| 16.2.2.1 | Protocol Deviations |
| 16.2.3 Patient | ts Excluded from the Efficacy Analysis |
| 16.2.3.1 | Subject Eligibility |
| 16.2.3.2 | Populations |
| 16.2.4 Demog | graphic Data |
| 16.2.4.1 | Demographic characteristics |
| 16.2.4.2 | History of GvHD |
| 16.2.4.3 | GvHD prophylaxis |
| 16.2.4.4 | Diagnostic of chronic GvHD |
| 16.2.4.5 | Ciclosporin therapy |
| 16.2.4.6 | Prednisone therapy |
| 16.2.4.7 | Concomitant treatments |
| | cy Response Data |
| 16.2.5.1 | Clinical assessment at each visit |
| 16.2.5.2 | Scores with abnormalities present but explained entirely by non-GVHD |
| 10.2.5.2 | documented cause at each visit |
| 16.2.5.3 | GvHD Chronic form A at each visit |
| 16.2.5.4 | Response at each visit |
| 16.2.6 Efficac | cy Response Data |
| 16.2.6.1 | All Adverse Events |
| 16.2.6.2 | Laboratory results |
| 16.2.6.3 | Physical examination |




### 17. APPENDICES

### 17.1 RESPONSE CALCULATION ALGORITHM

Etude GMED 16 001 : Evaluation des réponses complètes et partielles – 19/10/2020

Les réponses sont définies comme (règles de calcul basées sur le protocole et l'article Lee et al)

- Complete response at a visit: Lorsque tous les scores de « cGVDH activity assessment form A » des organes suivants sont à 0 ou que la variable "abnormalities present but explained entirely by non-GVHD documented cause » soit égale à Oui.

#### Détails :

Si une valeur est manquante pour un des organes atteints lors de la visite V1, la réponse ne peut pas être considérée comme complète. le fait que la valeur est manquante sera documentée.

Si une valeur à la visite d'intérêt est manquante sur un organe non atteint lors de la visite V1, la réponse complète peut être établie, car les réponses complètes ou partielles ne sont établies que sur les organes atteints à V1.

Si « abnormalities present but explained entirely by non-GVHD documented cause » = Oui pour un organe à la visite considérée, le score de cet organe n'est pas corrigé et cet organe n'est pas considéré pour l'évaluation de la réponse complète. cela ne créera pas de valeur manquante pour cet organe et n'empêchera pas la réponse d'être considérée comme complète si les informations sur les autres organes sont disponibles.

```
- BSA=0 ET skin features=0

M6_GVHD_A_S (préfixe M6 ou C1W6, W14, M9 et M12 selon la visite considérée)

M6_GVHD_A_S_F_S

M6_GVHD_A_S_ABN

- Eyes=0

M6_GVHD_A_E

M6_GVHD_A_E

M6_GVHD_A_E ABN
```

- Gastrointestinal=0 (pour chacun des 3 scores : Gastro-oesophageal, Gastro-upper, Gastro-lower) M6 GVHD A GASTRO1

```
M6_GVHD_A_GASTRO1
M6_GVHD_A_GASTRO3
M6_GVHD_GAST_ABN
```

- Mouth=0 (considérer la somme des 3 scores : Eythema, Lichenoid, Ulcers )

SAP-GvHD-ATO Study PASL201637-V3.0 Page 1987

Page 111 of 120




```
M6_GVHD_A_MOUTH1
M6_GVHD_A_MOUTH2
M6_GVHD_A_MOUTH3
M6_GVHD_MTH_ABN
```

Joint and fascia =0 M6\_GVHD\_A\_J M6\_GVHD\_A\_J\_ABN

Liver : les 3 valeurs (Bilirubine, ALAT et PAL) sont en dessous des ULN (Unité limite supérieure) si le score hépatique était >0 à V1 (table 1 et annexe du protocole)

Le score à V1 est calculé comme :

Score = 0: Bilirubine normale WITH ALAT AND PAL < 3 ULN

(.<V1\_GVHD\_A\_L\_BILI\_V<=V1\_GVHD\_A\_L\_BILI\_U\_V et
.<V1\_GVHD\_A\_L\_SGPT\_V<3\* V1\_GVHD\_A\_L\_SGPT\_U\_V et
.<V1\_GVHD\_A\_L\_ALK\_V<3\* V1\_GVHD\_A\_L\_ALK\_U\_V)

Score = 1 : Bilirubine normale WITH 3 ULN<=ALAT < 5 UNL AND 3 ULN <=PAL<5 UNL

Score = 2 : Bilirubine élevée (>1\*ULN) mais <= à 3 mg/dL OR ALAT >= 5 UNL OR PAL >=5 UNL (non mentionné dans article NIH).

Score = 3 : Bilirubine élevée > à 3 mg/dL

Lung : si FEV1 >= 80% et FEV1 < 70 à V1. et dans le cas où la valeur de FEV1 est manquante, si le score est égal à 0

```
M6_GVHD_A_LU_FEV1_V>= 80
missing(M6_GVHD_A_LU_FEV1_V) and M6_GVHD_A_L=0
M6_GVHD_A_L
M6_GVHD_A_L_ABN
```

Calcul de réponse par organe :

Aucun calcul de réponse par organe (complète, partielle ou progression) n'est effectué si :




- « abnormalities present but explained entirely by non-GVHD documented cause » = Oui pour un organe à la visite considérée
- CR\_organe, PR\_organe et PD\_organe sont alors mis à . (manquant)

Aucun calcul de réponse complète ou partielle par organe n'est effectué si :

- l'organe n'est pas atteint à V1 ou abnormalities present but explained entirely by non-GVHD documented cause » = Oui pour un organe à la visite V1.
- la progression est recherchée même si pas d'atteinte à V1
- CR\_organe et PR\_organe sont alors mis à . (manquant)
- **Partial response by organ**: en se basant sur les mêmes scores et en s'intéressant aux diminutions (ou augmentations) entre V1 (mêmes variables qu'indiquées précédemment mais qui commencent par « V1 » au lieu de « M6 ») et la visite considérée (M6,W6, W14, M9 ou M12)
- une diminution d'1 point pour les scores sur des échelles de 0 à 4 pour : Skin BSA, Skin features, Eyes, Joints, Gastro-oesophageal, Gastro-upper, Gastro-lower,
- une diminution de 2 points pour la somme des 3 sous-scores pour Mouth
- pour Lung, une augmentation entre V1 et la visite d'au moins 10% sur FEV1 avec FEV1 à V1 <70. Dans le cas de FEV1 manquants à V1 et ou M6, une diminution d'1 point sur le score 'lungs'
- pour Liver, (Bilirubine, ALAT ou PAL),
- si les valeurs à M6 sont en dessous des normales, la réponse est considérée Complète
- sinon la recherche d'une réponse partielle est effectuée : diminution de 50% de la valeur initiale Le ratio est calculé ainsi : (M6-V1/V1)\*100 et si le ratio est inférieur à -50 (mais pas de progression pour une des autres valeurs), il y a une réponse partielle

Global Partial response: au moins une réponse partielle sur un organe et avec une absence de progression pour un autre site

- Progressive disease by organ:
- peau, yeux, œsophage, tractus gastro-intestinal supérieur et inférieur : augmentation 1 point ou plus sur échelle de 0 à 3 = progression *SAUF* si changement de 0 à 1 (progression non spécifique)
- Joint: augmentation d'1 point ou plus = progression
- bouche : changement de 2 points ou plus sur la somme des 3 sous-scores




- pour Lung, diminution de 10 % avec FEV1 à V1 < 75% . Dans le cas de FEV1 manquants, augmentation d'1 point ou plus SAUF si changement de 0 à 1 (progression non spécifique)
- pour Liver, si l'une des valeurs à M6 est au-dessus de la normale pour Bilirubine, ALAT ou PAL, la recherche d'une progression est effectuée : la différence M6-V1 est calculée et si la différence est supérieure à 2\*ULN, il y a Progression.

Global progressive disease: si au moins un site avec une progression

Mixed response: si Progressive disease sur au moins un organe et Partial response sur au moins un autre

### Extraits du protocole :

Table 4. Response determination for chronic GvHD (extrait du protocole)

| Organ | Complete Response | Partial Response | Progression |
|---|---|---|---|
| Skin | NIH Skin Score 0 after | Decrease in NIH Skin Score | Increase in NIH Skin Score by 1 or |
| | previous involvement | by 1 or more points | more points, except 0 to 1 |
| Eyes | NIH Eye Score 0 after | Decrease in NIH Eye Score | Increase in NIH Eye Score by 1 or |
| | previous involvement | by 1 or more points | more points, except 0 to 1 |
| Mouth | NIH Modified OMRS 0 after | Decrease in NIH Modified OMRS | Increase in NIH Modified OMRS |
| | previous involvement | of 2 or more points | of 2 or more points |
| Esophagus | NIH Esophagus Score 0 after | Decrease in NIH Esophagus | Increase in NIH Esophagus Score |
| | previous involvement | Score by 1 or more points | by 1 or more points, except 0 to 1 |
| Upper GI | NIH Upper GI Score 0 after | Decrease in NIH Upper GI | Increase in NIH Upper GI Score |
| | previous involvement | Score by 1 or more points | by 1 or more points, except 0 to 1 |
| Lower GI | NIH Lower GI Score 0 after | Decrease in NIH Lower GI | Increase in NIH Lower GI Score by 1 |
| | previous involvement | Score by 1 or more points | or more points, except from 0 to 1 |
| Liver | Normal ALT, alkaline | Decrease by 50% | Increase by $2 \times ULN$ |
| | phosphatase, and Total | | - |
| | bilirubin after previous | | |
| | elevation of 1 or more | | |
| Lungs | - Normal %FEV1 after | <ul> <li>Increase by 10% predicted</li> </ul> | - Decrease by 10% predicted |
| | previous involvement | absolute value of %FEV1 | absolute value of %FEV1 |
| | - If PFTs not available, NIH | <ul> <li>If PFTs not available, decrease</li> </ul> | - If PFTs not available, increase in |
| | Lung Symptom Score 0 | in NIH Lung Symptom Score | NIH Lung Symptom Score by 1 |
| | after previous involvement | by 1 or more points | or more points, except 0 to 1 |
| Joints and fascia | Both NIH Joint and Fascia | Decrease in NIH Joint and Fascia | Increase in NIH Joint and Fascia |
| | Score 0 and P-ROM score | Score by 1 or more points or | Score by 1 or more points or |
| | 25 after previous involvement | increase in P-ROM score by 1 | decrease in P-ROM score by 1 |
| | by at least 1 measure | point for any site | point for any site |
| Global | Clinician overall severity score 0 | Clinician overall severity score | Clinician overall severity score |
| | _ | decreases by 2 or more points | increases by 2 or more points |
| | | on a 0-10 scale | on a 0-10 scale |

ULN indicates upper limit of normal.




# Appendix 2: Organ scoring of cGvHD

(NIH consensus criteria, Jagasia et al. Bone Marrow Transplant, 2015)

| | SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
|---|---|---|---|---|
| EYES Keratoconjunctivitis sicca (KCS) confirmed by ophthalmologist: Yes No Not examined | □ No symptoms | ☐ Mild dry eye symptoms not affecting ADL (requirement of lubricant eye drops ≤ 3 x per day) | □ Moderate dry eye symptoms partially affecting ADL (requiring lubricant eye drops > 3 x per day or punctal plugs), WITHOUT new vision impairment due to KCS | affecting ADL (special |
| | на ехриитей етигету в | by non-GVHD documente | eu cuuse (specijy): | |
| GI Tract Check all that apply: Esophageal web/ proximal stricture or ring Dysphagia Anorexia Nausea Vomiting Diarrhea Weight loss >5%* Failure to thrive Abnormality present by | □ No symptoms out explained entirely | Symptoms without significant weight loss* (<5%) | Symptoms associated with mild to moderate weight loss* (5-15%) OR moderate diarrhea without significant interference with daily living | □ Symptoms associated with significant weight loss* >15%, requires nutritional supplement for most calorie needs OR esophageal dilation OR severe diarrhea with significant interference with daily living |
| LIVER | ☐ Normal total<br>bilirubin and<br>ALT or AP<br>< 3 x ULN | □ Normal total bilirubin with ALT ≥3 to 5 x ULN or AP > 3 x ULN | ☐ Elevated total<br>bilirubin but<br>≤3 mg/dL or<br>ALT > 5 ULN | ☐ Elevated total<br>bilirubin > 3 mg/dL |
| ☐ Abnormality present b | out explained entirely | by non-GVHD documente | ed cause (specify): | |
| Lungs** | | | | |
| Symptom score: | □ No symptoms | ☐ Mild symptoms<br>(shortness of<br>breath after<br>climbing one flight<br>of steps) | ☐ Moderate<br>symptoms<br>(shortness of breath<br>after walking on<br>flat ground) | $\square$ Severe symptoms<br>(shortness of breath at rest; requiring $0_2$ ) |
| Lung score: % FEV1 | □ FEV1≥80% | □ FEV1 60-79% | □ FEV1 40-59% | □ FEV1 ≤39% |
| Pulmonary function tests Not performed | | by non-GVHD documente | ad agusa (anaaifu): | |
| □ Abnormanty present b | на ехрииней епигету г | оу пон-Өүнэ аоситепи | a cause (specify): | |


## 17.2 FACT-BMT

## 17.2.1 FACT-BMT items

#### FACT-BMT (4ème Version)

Veuillez indiquer votre réponse en entourant un seul chiffre par ligne et en tenant compte des  $\underline{7~derniers~jours}$ .

| | <u>AUTRES SUJETS D'INQUIÉTUDE</u> | Pas du<br>tout | Un<br>peu | Moyen-<br>nement | Beau-<br>coup | Énormé-<br>ment |
|---|---|---|---|---|---|---|
| BMT1 | Je m'inquiète de ne pas pouvoir continuer à travailler (y compris le travail à la maison) | 0 | 1 | 2 | 3 | 4 |
| BMT2 | Je me sens distant(e) des autres | 0 | 1 | 2 | 3 | 4 |
| вмт3 | J'ai peur que la greffe ne réussisse pas | 0 | 1 | 2 | 3 | 4 |
| BMT4 | Les effets du traitement sont pires que ce que j'imaginais | 0 | 1 | 2 | 3 | 4 |
| C6 | J'ai bon appétit | 0 | 1 | 2 | 3 | 4 |
| C7 | Je suis satisfait(e) de mon apparence physique | 0 | 1 | 2 | 3 | 4 |
| BMT5 | Je peux me débrouiller seul(e) | 0 | 1 | 2 | 3 | 4 |
| вмт6 | Je me fatigue facilement | 0 | 1 | 2 | 3 | 4 |
| BL4 | Le sexe m'intéresse | 0 | 1 | 2 | 3 | 4 |
| BMT7 | J'ai peur de ne plus pouvoir avoir d'enfants | 0 | 1 | 2 | 3 | 4 |
| BMT8 | J'ai confiance en mes infirmières(iers) | 0 | 1 | 2 | 3 | 4 |
| вмт9 | Je regrette d'avoir eu une greffe de la moelle osseuse | 0 | 1 | 2 | 3 | 4 |
| BMT<br>10 | J'ai de la mémoire | 0 | 1 | 2 | 3 | 4 |
| Br1 | Je suis capable de me concentrer | 0 | 1 | 2 | 3 | 4 |
| BMT<br>11 | J'ai fréquemment des rhumes ou des infections | 0 | 1 | 2 | 3 | 4 |
| BMT<br>12 | Je vois trouble | 0 | 1 | 2 | 3 | 4 |
| BMT<br>13 | Je suis gêné(e) par un changement de goût des aliments | 0 | 1 | 2 | 3 | 4 |
| BMT<br>14 | J'ai des tremblements | 0 | 1 | 2 | 3 | 4 |
| В1 | J'ai le souffle court | 0 | 1 | 2 | 3 | 4 |
| BMT<br>15 | Je suis gêné(e) par des problèmes de peau (éruptions démangeaisons) | 0 | 1 | 2 | 3 | 4 |
| BMT<br>16 | J'ai du mal à aller à la selle | 0 | 1 | 2 | 3 | 4 |
| BMT<br>17 | Ma maladie est une lourde épreuve pour ma famille proche | 0 | 1 | 2 | 3 | 4 |
| BMT<br>18 | Le coût du traitement est un fardeau pour moi et pour ma famille | 0 | 1 | 2 | 3 | 4 |

17 February 2010: 17 February 2010: 17 February 2010: 18 February




#### FACT-BMT (4ème Version)

Vous trouverez ci-dessous une liste de commentaires que d'autres personnes atteintes de la même maladie que vous ont jugés importants. **Veuillez indiquer votre réponse en entourant un seul chiffre par ligne et en tenant compte des <u>7 derniers jours</u>.** 

| | BIEN-ÊTRE PHYSIQUE | Pas du<br>tout | Un<br>peu | Moyen-<br>nement | Beau-<br>coup | Énormé-<br>ment |
|---|---|---|---|---|---|---|
| GP1 | Je manque d'énergie | 0 | 1 | 2 | 3 | 4 |
| GP2 | J'ai des nausées | 0 | 1 | 2 | 3 | 4 |
| GP3 | À cause de mon état physique, j'ai du mal à répondre aux besoins de ma famille | 0 | 1 | 2 | 3 | 4 |
| GP4 | J'ai des douleurs | 0 | 1 | 2 | 3 | 4 |
| GP5 | Je suis incommodé(e) par les effets secondaires du traitement | 0 | 1 | 2 | 3 | 4 |
| GP6 | Je me sens malade | 0 | 1 | 2 | 3 | 4 |
| GP7 | Je suis obligé(e) de passer du temps allongé(e) | 0 | 1 | 2 | 3 | 4 |
| | BIEN-ÊTRE FAMILIAL/SOCIAL | Pas du tout | Un<br>peu | Moyen-<br>nement | Beau-<br>coup | Énormé-<br>ment |
| GS1 | Je me sens proche de mes amis | 0 | 1 | 2 | 3 | 4 |
| GS2 | Ma famille me soutient moralement | 0 | 1 | 2 | 3 | 4 |
| GS3 | Mes amis me soutiennent | 0 | 1 | 2 | 3 | 4 |
| GS4 | Ma famille a accepté ma maladie | . 0 | 1 | 2 | 3 | 4 |
| GS5 | Je suis satisfait(e) de la communication avec ma famille au sujet de ma maladie | 0 | 1 | 2 | 3 | 4 |
| GS6 | Je me sens proche de mon (ma) partenaire (ou de la personne qui est mon principal soutien) | 0 | 1 | 2 | 3 | 4 |
| Q1 | Quel que soit votre degré d'activité sexuelle en ce<br>moment, veuillez répondre à la question suivante.<br>Si vous préférez ne pas y répondre, cochez cette case<br>et passez à la section suivante. | | | | | |
| GS7 | Je suis satisfait(e) de ma vie sexuelle | 0 | 1 | 2 | 3 | 4 |

 French (Universal)
 17 February 2010

 Copyright 1987, 1997
 Page 1 of 3




#### FACT-BMT (4ème Version)

Veuillez indiquer votre réponse en entourant un seul chiffre par ligne et en tenant compte des 7 derniers jours.

| | BIEN-ÊTRE ÉMOTIONNEL | Pas du<br>tout | Un<br>peu | Moyen-<br>nement | Beau-<br>coup | Énormé-<br>ment |
|---|---|---|---|---|---|---|
| GE1 | Je me sens triste | 0 | 1 | 2 | 3 | 4 |
| GE2 | Je suis satisfait(e) de la façon dont je fais face à ma<br>maladie | 0 | 1 | 2 | 3 | 4 |
| GE3 | Je perds espoir dans le combat contre ma maladie | 0 | 1 | 2 | 3 | 4 |
| GE4 | Je me sens nerveux (nerveuse) | 0 | 1 | 2 | 3 | 4 |
| GE5 | Je suis préoccupé(e) par l'idée de mourir | 0 | 1 | 2 | 3 | 4 |
| GE6 | Je suis préoccupé(e) à l'idée que mon état de santé<br>puisse s'aggraver | 0 | 1 | 2 | 3 | 4 |
| | BIEN-ÊTRE FONCTIONNEL | Pas du<br>tout | Un<br>peu | Moyen-<br>nement | Beau-<br>coup | Énormé-<br>ment |
| GF1 | BIEN-ÊTRE FONCTIONNEL Je suis capable de travailler (y compris le travail à la maison) | | | | | |
| GF1 | Je suis capable de travailler (y compris le travail | tout | peu | nement | coup | ment |
| | Je suis capable de travailler (y compris le travail à la maison) | 0 | peu<br>1 | nement 2 | coup 3 | ment 4 |
| GF2 | Je suis capable de travailler (y compris le travail à la maison) | 0 | peu 1 | nement 2 2 | 3<br>3 | ment 4 |
| GF2<br>GF3 | Je suis capable de travailler (y compris le travail à la maison) Mon travail (y compris le travail à la maison) me donne de la satisfaction | 0<br>0<br>0 | peu 1 1 1 1 1 | nement 2 2 2 | 3<br>3<br>3 | 4 4 4 |
| GF2<br>GF3 | Je suis capable de travailler (y compris le travail à la maison) Mon travail (y compris le travail à la maison) me donne de la satisfaction Je suis capable de profiter de la vie J'ai accepté ma maladie | 0<br>0<br>0<br>0 | peu 1 1 1 1 | 2 2 2 2 2 | 3 3 3 3 | 4 4 4 4 |

French (Universal) 17 February 20

## 17.2.2 Details of FACT-BMT calculation






## 17.3 LEE SYMPTOM SCALE

The Lee Chronic GVHD Symptom Scale is a 30 item instrument with 7 subscales (skin, eyes, mouth, lung, nutrition, energy and psych) containing 2-7 items. Response options for "let us know if you have been bothered by any of the following in the past month" range from 0-4 (Not at all, Slightly, Moderately, Quite a bit, Extremely). Some investigators have used the scale in reference to the past 7 days. (Lee SJ, Cook EF, Soiffer R, Antin JH. Development and validation of a scale to measure symptoms of chronic graft-versus-host disease. *Biol Blood Marrow Transplant* 2002; 8:444-452)

| Subscale name | Number of items | Items |
|---|---|---|
| Skin | 5 | a. Abnormal skin color |
| | | b. Rashes |
| | | c. Thickened skin |
| | | d. Sores on skin |
| | | e. Itchy skin |
| Eye | 3 | f. Dry eyes |
| | | g. Need to use eyedrops frequently |
| | | h. Difficulty seeing clearly |
| Mouth | 2 | i. Need to avoid certain foods due to mouth pain |
| | | j. Ulcers in mouth |
| Lung | 5 | I. Frequent cough |
| | | m. Colored sputum |
| | | o. Shortness of breath at rest |
| | | p. Need to use oxygen |
| | | aa. Fevers |
| Nutrition | 5 | k. Receiving nutrition from an intravenous line or feeding tube |




| | | q. Difficulty swallowing solid foods |
|--------|---|--------------------------------------|
| | | r. Difficulty swallowing liquids |
| | | s. Vomiting |
| | | t. Weight loss |
| Energy | 7 | n. Shortness of breath with exercise |
| | | u. Joint and muscle aches |
| | | v. Limited joint movement |
| | | w. Muscle cramps |
| | | x. Weak muscles |
| | | y. Loss of energy |
| | | z. Need to sleep more/take naps |
| Psych | 3 | bb. Depression |
| | | cc. Anxiety |
| | | dd. Difficulty sleeping |

**Bold** indicates items that are scored under a different subscale than where they are located

#### Scoring rules:

- 1. Note that the subscales do not conform exactly to the categories in the patient survey.
- 2. Subscales may be scored if 50% of more of the items in the subscale are completed.
- 3. Scores are linearly transformed to a 0-100 scale where 0 means all answered items were a "0" and "100" means that all answered items were a "4"
- 4. Missing items are not included in the scoring.
- 5. The summary score is the average of the subscale scores, as long as 4 or more subscales are available.
- 6. Higher scores indicate more severe symptoms.
  - 7. A clinically meaningful difference for each subscale or the summary score is considered to be half a standard deviation of the baseline score for the population, based on the distribution method of determining clinically meaningful changes.